CLINICAL TRIAL: NCT03963401
Title: A PHASE 2B, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY OF PF-06700841 TO EVALUATE THE EFFICACY AT 16 WEEKS AND TO EVALUATE THE SAFETY AND EFFICACY UP TO 1 YEAR IN SUBJECTS WITH ACTIVE PSORIATIC ARTHRITIS
Brief Title: A Study to Evaluate the Efficacy and Safety of PF-06700841 in Subjects With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7931030; 2018-004241-16 (EudraCT Number)
Record Dates: First submitted 2019-05-15; First posted 2019-05-24 (Actual); Results first posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Psoriatic Arthritis
Keywords: Spondyloarthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Spondylarthritis | interventions — PF-06700841

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- PF-06700841 60 mg once daily (Experimental): PF-06700841 60 mg once daily for 52 weeks
  Interventions: Drug: PF-06700841
- PF-06700841 30 mg once daily (Experimental): PF-06700841 30 mg once daily for 52 weeks
  Interventions: Drug: PF-06700841
- PF-06700841 10 mg once daily followed by 60 mg once daily (Experimental): PF-06700841 10 mg once daily for 16 weeks, followed by 60 mg once daily until Week 52
  Interventions: Drug: PF-06700841
- PF-06700841 10 mg once daily followed by 30 mg once daily (Experimental): PF-06700841 10 mg once daily for 16 weeks, followed by 30 mg once daily until Week 52
  Interventions: Drug: PF-06700841
- Placebo once daily followed by 60 mg once daily (Placebo Comparator): Placebo once daily for 16 weeks, followed by PF-06700841 60 mg once daily until Week 52
  Interventions: Other: Placebo
- Placebo once daily followed by 30 mg once daily (Placebo Comparator): Placebo once daily for 16 weeks, followed by PF-06700841 30 mg once daily until Week 52
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-06700841 — Starting after the Week 16 visit, subjects receiving PF-06700841 10 mg once daily will start to randomly receive either the 60 mg QD dose or 30 mg QD dose until Week 52, as predetermined at randomization. All subjects will receive blinded dosing throughout the 52 weeks study treatment period in order to maintain the study blind.
  Arms: PF-06700841 10 mg once daily followed by 30 mg once daily; PF-06700841 10 mg once daily followed by 60 mg once daily; PF-06700841 30 mg once daily; PF-06700841 60 mg once daily
Other: Placebo — Starting after the Week 16 visit, subjects receiving placebo will start to randomly receive either the 60 mg QD dose or 30 mg QD dose until Week 52, as predetermined at randomization. All subjects will receive blinded dosing throughout the 52 weeks study treatment period in order to maintain the study blind.
  Arms: Placebo once daily followed by 30 mg once daily; Placebo once daily followed by 60 mg once daily

SUMMARY:
This is a 52 week Phase 2b study designed to evaluate the efficacy at 16 weeks and to evaluate the safety and efficacy up to 1 year in subjects with active psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Active arthritis at screening/baseline as indicated by >/= 3 tender/painful and 3 swollen joints.
* Active plaque psoriasis at screening and baseline.

Exclusion Criteria:

* Non-plaque forms of psoriasis (with exception of nail psoriasis).
* History of autoimmune rheumatic disease other than PsA; also prior history of or current, rheumatic inflammatory disease other than PsA.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- Australia (2):
  - Rheumatology Research Unit, Maroochydore, Queensland
  - Emeritus Research, Melbourne, Victoria
- Bulgaria (6):
  - MHAT Trimontium OOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment "Pulmed", Plovdiv
  - University Multiprofile Hospital for Active Treatment ''Plovdiv'' AD, Plovdiv
  - Medical Center "Pirogov", Sofia
  - "Diagnostic-Consulting Center XVII - Sofia", Sofia
  - University Multiprofile Hospital for Active Treatment Sveti Ivan Rilski, Sofia
- Czechia (5):
  - L.K.N. Arthrocentrum s.r.o., Hlučín
  - CCR Czech a.s., Pardubice
  - Revmatologicky ustav, Prague
  - CCR Prague s.r.o., Prague
  - MEDICAL PLUS s.r.o., Uherské Hradiště
- Estonia (3):
  - Innomedica OU, Tallinn
  - Center for Clinical and Basic Research, Tallinn
  - East Tallinn Central Hospital, Tallinn
- Hungary (2):
  - Qualiclinic Kft., Budapest
  - VITAL MEDICAL CENTER Orvosi es Fogorvosi Kozpont, Veszprém
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences, Kauno klinikos, Kaunas
  - National Osteoporosis Center, Vilnius
- Poland (10):
  - ZDROWIE Osteo-Medic s.c. L. I A. Racewicz, A. i J. Supronik, Bialystok
  - ClinicMed Daniluk Nowak Sp. Jawna, Bialystok
  - Zespol Poradni Specjalistycznych "REUMED" Filia nr 2, Lublin
  - NZOZ Lecznica Mak-Med s.c., Nadarzyn
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Ai Centrum Medyczne Sp. z o.o. Sp. k., Poznan
  - Prywatna Praktyka Lekarska Prof. UM dr hab. med. Pawel Hrycaj, Poznan
  - RCMed Oddzial Sochaczew, Sochaczew
  - NASZ LEKARZ Przychodnie Medyczne, Torun
  - REUMATIKA - Centrum Reumatologii NZOZ, Warsaw
- Russia (10):
  - LLC "Family Outpatient clinic #4", Korolyov, Moscow Oblast
  - FGBOU VO "Orenburg State Medical University" of the Ministry of Health of the Russian Federation, Orenburg
  - GBUZ "Orenburg Regional Clinical Hospital", Orenburg
  - SBHI of the Republic of Karelia "Republican Hospital n. a. V.A. Baranov", Petrozavodsk
  - FSBEI of HE "Ryazan State Medical University n. a academician I.P.Pavlov", Ryazan
  - SBI of Ryazan Region "Regional Clinical Hospital", Ryazan
  - Limited Liability Company "Sanavita", Saint Petersburg
  - GUZ "Regional Clinical Hospital", Saratov
  - LLC "BioMed", Vladimir
  - State Autonomous Healthcare Institution of Yaroslavl Region, Yaroslavl
- Serbia (2):
  - Institute of Rheumatology, Belgrade
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
- Slovakia (3):
  - Narodny ustav reumatickych chorob, Piešťany
  - MUDr. Zuzana Cizmarikova, s.r.o., Poprad
  - REUMEX s.r.o., Rimavská Sobota
- Spain (3):
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitario A Coruna, A Coruña
  - Hospital Quironsalud Infanta Luisa, Seville

REFERENCES:
- [Background] Banfield C, Scaramozza M, Zhang W, Kieras E, Page KM, Fensome A, Vincent M, Dowty ME, Goteti K, Winkle PJ, Peeva E. The Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a TYK2/JAK1 Inhibitor (PF-06700841) in Healthy Subjects and Patients With Plaque Psoriasis. J Clin Pharmacol. 2018 Apr;58(4):434-447. doi: 10.1002/jcph.1046. Epub 2017 Dec 21. PMID 29266308
- [Derived] Mease P, Helliwell P, Silwinska-Stanczyk P, Miakisz M, Ostor A, Peeva E, Vincent MS, Sun Q, Sikirica V, Winnette R, Qiu R, Li G, Feng G, Beebe JS, Martin DA. Efficacy and Safety of the TYK2/JAK1 Inhibitor Brepocitinib for Active Psoriatic Arthritis: A Phase IIb Randomized Controlled Trial. Arthritis Rheumatol. 2023 Aug;75(8):1370-1380. doi: 10.1002/art.42519. Epub 2023 Jun 22. PMID 37194394
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7931030

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 219 participants were enrolled in this study and 1 of them didn't receive any study treatment.
Groups:
- PF-06700841 60 mg QD -> PF-06700841 60 mg QD: PF-06700841 tablet was administered orally at 60 milligram (mg) once daily (QD) during both the initial period (from Day 1 to Week 16) and the extension period (Week 17 through Week 52).
- PF-06700841 30 mg QD -> PF-06700841 30 mg QD: PF-06700841 tablet was administered orally at 30 mg QD during both the initial period (from Day 1 to Week 16) and the extension period (Week 17 through Week 52).
- PF-06700841 10 mg QD -> PF-06700841 60 mg QD: PF-06700841 tablet was administered orally at 10 mg QD during the initial period (from Day 1 to Week 16) and PF-06700841 tablet was administered orally at 60 mg QD during the extension period (Week 17 through Week 52).
- PF-06700841 10 mg QD -> PF-06700841 30 mg QD: PF-06700841 tablet was administered orally at 10 mg QD during the initial period (from Day 1 to Week 16) and PF-06700841 tablet was administered orally at 30 mg QD during the extension period (Week 17 through Week 52).
- Placebo -> PF-06700841 60 mg QD: Placebo matched to PF-06700841 tablet was administered orally QD during the initial period (from Day 1 to Week 16) and PF-06700841 tablet was administered orally at 60 mg during the extension period (Week 17 through Week 52).
- Placebo -> PF-06700841 30 mg QD: Placebo matched to PF-06700841 tablet was administered orally QD during the initial period (from Day 1 to Week 16) and PF-06700841 tablet was administered orally at 30 mg during the extension period (Week 17 through Week 52).
Period: Initial Period (Day 1 - Week 16)
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Started | 60 | 61 | 16 | 15 | 34 | 33
Treated | 60 | 60 | 16 | 15 | 34 | 33
Completed | 57 | 57 | 14 | 13 | 31 | 31
Not Completed | 3 | 4 | 2 | 2 | 3 | 2
Not completed — Adverse Event | 1 | 2 | 0 | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1 | 2 | 0
Not completed — Randomized but Not Treated | 0 | 1 | 0 | 0 | 0 | 0
Period: Extension Period (Week 17 - Week 52)
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Started | 57 | 57 | 14 | 13 | 31 | 31
Completed | 43 | 52 | 10 | 12 | 25 | 26
Not Completed | 14 | 5 | 4 | 1 | 6 | 5
Not completed — Adverse Event | 6 | 3 | 2 | 0 | 4 | 3
Not completed — Lack of Efficacy | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Non-Compliance With Study Drug | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 0 | 1 | 1
Not completed — No Longer Meets Eligibility Criteria | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were randomized to the study and received at least one dose of the randomized study treatment.
Groups:
- PF-06700841 60 mg QD -> PF-06700841 60 mg QD: PF-06700841 tablet was administered orally at 60 mg once daily (QD) during both the initial period (from Day 1 to Week 16) and the extension period (Week 17 through Week 52).
- Total: Total of all reporting groups
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD | Total
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33 | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.7 (11.47) | 45.9 (10.23) | 47.8 (14.16) | 47.7 (12.95) | 47.9 (12.58) | 48.5 (11.84) | 47.6 (11.62)
Age, Continuous [Median (Full Range); unit: Years] | 50.0 [24 to 70] | 46.0 [26 to 73] | 43.5 [22 to 71] | 47.0 [28 to 73] | 48.0 [21 to 69] | 50.0 [23 to 72] | 48.0 [21 to 73]
Age, Customized [Number; unit: Participants]
  18-44 | 22 | 26 | 9 | 6 | 13 | 14 | 90
  45-64 | 35 | 31 | 5 | 8 | 17 | 16 | 112
  ≥65 | 3 | 3 | 2 | 1 | 4 | 3 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 7 | 7 | 20 | 16 | 116
  Male | 26 | 28 | 9 | 8 | 14 | 17 | 102
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 59 | 60 | 16 | 15 | 34 | 33 | 217
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 60 | 59 | 16 | 15 | 33 | 32 | 215
  Not reported | 0 | 1 | 0 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an American College of Rheumatology 20 (ACR20) Response at Week 16
Description: ACR 20 was calculated as a ≥20% improvement in tender and swollen joint counts and ≥20% improvement in 3 of the 5 remaining ACR core set measures: patient pain assessment (a horizontal visual analog scale assessment of the patient's level of pain), patient global assessment (the patient's overall assessment of how the arthritis was doing by a visual analog scale), physician global assessment (a horizontal visual analog scale measure of the physician's assessment of the patient's current disease activity), patient self-assessed disability (a validated and reliable patient self-assessment instrument which measured physical functions in rheumatoid arthritis patients) and an acute-phase reactant (C-reactive protein level). The participants receiving placebo in the initial period (Day 1 - Week 16) were combined into a single placebo group, while those who received PF-06700841 (10 mg QD) in the initial period were combined into a single PF-06700841 10 mg QD group.
Time Frame: Week 16
Population: All participants who received at least 1 dose of the randomized study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Placebo: Placebo matched to PF-06700841 tablet was administered orally QD during the initial period (from Day 1 to Week 16).
- PF-06700841 10 mg QD: PF-06700841 tablet was administered orally at 10 mg QD during the initial period (from Day 1 to Week 16).
- PF-06700841 30 mg QD: PF-06700841 tablet was administered orally at 30 mg QD during the initial period (from Day 1 to Week 16).
- PF-06700841 60 mg QD: PF-06700841 tablet was administered orally at 60 mg QD during the initial period (from Day 1 to Week 16).
Arm/Group | Placebo | PF-06700841 10 mg QD | PF-06700841 30 mg QD | PF-06700841 60 mg QD
Number analyzed (Participants) | 67 | 31 | 60 | 59
Percentage of participants | 43.28 [31.42 to 55.15] | 64.52 [47.67 to 81.36] | 66.67 [54.74 to 78.59] | 74.58 [63.47 to 85.69]
Statistical Analysis 1: Comparison: Placebo vs PF-06700841 10 mg QD; Test type: Superiority; p = 0.1172, Normal approximation, Dunnett's method; Mean Difference (Final Values) = 21.23, 90% CI 2-sided [3.94 to 38.52], Standard Error of Mean 10.51
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 30 mg QD; Test type: Superiority; p = 0.0197, Normal approximation, Dunnett's Method; Median Difference (Final Values) = 23.38, 90% CI 2-sided [9.26 to 37.50], Standard Error of Mean 8.58
Statistical Analysis 3: Comparison: Placebo vs PF-06700841 60 mg QD; Test type: Superiority; p = 0.0006, Normal approximation, Dunnett's Method; Median Difference (Final Values) = 31.29, 90% CI 2-sided [17.65 to 44.93], Standard Error of Mean 8.29

2. Secondary Outcome: Percentage of Participants Achieving an ACR20 Response at Week 16 in the Subgroup of Participants Who Were Tumor Necrosis Factor (TNF) α Inhibitor naïve
Description: as for outcome 1
Time Frame: Week 16
Population: All participants who received at least 1 dose of the randomized study treatment with prior TNFα naïve.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06700841 10 mg QD | PF-06700841 30 mg QD | PF-06700841 60 mg QD
Number analyzed (Participants) | 60 | 28 | 56 | 55
Percentage of participants | 43.33 [30.79 to 55.87] | 64.29 [46.54 to 82.03] | 69.64 [57.60 to 81.69] | 74.55 [63.03 to 86.06]
Statistical Analysis 1: Comparison: Placebo vs PF-06700841 10 mg QD; Test type: Superiority; p = 0.0588, Normal approximation method; Mean Difference (Final Values) = 20.95, 90% CI 2-sided [2.72 to 39.19], Standard Error of Mean 11.09
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 30 mg QD; Test type: Superiority; p = 0.0030, Normal approximation method; Median Difference (Final Values) = 26.31, 90% CI 2-sided [11.72 to 40.90], Standard Error of Mean 8.87
Statistical Analysis 3: Comparison: Placebo vs PF-06700841 60 mg QD; Test type: Superiority; p = 0.0003, Normal approximation method; Median Difference (Final Values) = 31.21, 90% CI 2-sided [16.93 to 45.50], Standard Error of Mean 8.68

3. Secondary Outcome: Percentage of Participants Achieving an ACR20 Response at Weeks 2, 4, 8, 12, 20, 28, 36, 44 and 52
Description: The American College of Rheumatology's definition for calculating improvement in rheumatoid arthritis (ACR20) was calculated as a ≥20% improvement in tender and swollen joint counts and ≥20% improvement in 3 of the 5 remaining ACR core set measures: patient pain assessment (a horizontal visual analog scale assessment of the patient's level of pain), patient global assessment (the patient's overall assessment of how the arthritis was doing by a visual analog scale), physician global assessment (a horizontal visual analog scale measure of the physician's assessment of the patient's current disease activity), patient self-assessed disability (a validated and reliable patient self-assessment instrument which measured physical functions in rheumatoid arthritis patients) and an acute-phase reactant (C-reactive protein level).
Time Frame: Weeks 2, 4, 8, 12, 20, 28, 36, 44 and 52
Population: All participants who received at least 1 dose of the randomized study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PF-06700841 10 mg QD -> PF-06700841 60 mg QD: PF-06700841 tablet was administered orally at 10 mg QD from Day 1 to Week 16. From Week 17 to Week 52, PF-06700841 tablet was administered orally at 60 mg QD.
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Percentage of participants
  Week 2 | 21.67 [11.24 to 32.09] | 18.33 [8.54 to 28.12] | 18.75 [0.00 to 37.87] | 3.13 [0.00 to 11.65] | 5.88 [0.00 to 13.79] | 18.18 [5.02 to 31.34]
  Week 4 | 45.00 [32.41 to 57.59] | 51.67 [39.02 to 64.31] | 31.25 [8.54 to 53.96] | 20.00 [0.00 to 40.24] | 14.71 [2.80 to 26.61] | 24.24 [9.62 to 38.86]
  Week 8 | 66.67 [54.74 to 78.59] | 55.00 [42.41 to 67.59] | 50.00 [25.50 to 74.50] | 40.00 [15.21 to 64.79] | 35.29 [19.23 to 51.36] | 42.42 [25.56 to 59.29]
  Week 12 | 70.00 [58.40 to 81.60] | 63.33 [51.14 to 75.53] | 56.25 [31.94 to 80.56] | 60.00 [35.21 to 84.79] | 44.12 [27.43 to 60.81] | 39.39 [22.72 to 56.07]
  Week 20 | 81.67 [71.88 to 91.46] | 80.00 [69.88 to 90.12] | 68.75 [46.04 to 91.46] | 60.00 [35.21 to 84.79] | 73.53 [58.70 to 88.36] | 75.76 [61.14 to 90.38]
  Week 28 | 73.33 [62.14 to 84.52] | 78.33 [67.91 to 88.76] | 68.75 [46.04 to 91.46] | 73.33 [50.95 to 95.71] | 64.71 [48.64 to 80.77] | 81.82 [68.66 to 94.98]
  Week 36 | 66.67 [54.74 to 78.59] | 78.33 [67.91 to 88.76] | 68.75 [46.04 to 91.46] | 80.00 [59.76 to 100.00] | 64.71 [48.64 to 80.77] | 81.82 [68.66 to 94.98]
  Week 44 | 68.33 [56.56 to 80.10] | 73.33 [62.14 to 84.52] | 62.50 [38.78 to 86.22] | 73.33 [50.95 to 95.71] | 67.65 [51.92 to 83.37] | 75.76 [61.14 to 90.38]
  Week 52 | 61.67 [49.36 to 73.97] | 70.00 [58.40 to 81.60] | 56.25 [31.94 to 80.56] | 60.00 [35.21 to 84.79] | 61.76 [45.43 to 78.10] | 66.67 [50.58 to 82.75]

4. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The American College of Rheumatology's definition for calculating improvement in rheumatoid arthritis (ACR50) was calculated as a ≥50% improvement in tender and swollen joint counts and ≥50% improvement in 3 of the 5 remaining ACR core set measures: patient pain assessment (a horizontal visual analog scale assessment of the patient's level of pain), patient global assessment (the patient's overall assessment of how the arthritis was doing by a visual analog scale), physician global assessment (a horizontal visual analog scale measure of the physician's assessment of the patient's current disease activity), patient self-assessed disability (a validated and reliable patient self-assessment instrument which measured physical functions in rheumatoid arthritis patients) and an acute-phase reactant (C-reactive protein level).
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: All participants who received at least 1 dose of the randomized study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Percentage of participants
  Week 2 | 6.67 [0.35 to 12.98] | 1.67 [0.00 to 4.91] | 2.94 [0.00 to 10.97] | 3.13 [0.00 to 11.65] | 1.43 [0.00 to 5.36] | 1.47 [0.00 to 5.52]
  Week 4 | 13.33 [4.73 to 21.93] | 16.67 [7.24 to 26.10] | 2.94 [0.00 to 10.97] | 6.67 [0.00 to 19.29] | 2.94 [0.00 to 8.62] | 6.06 [0.00 to 14.20]
  Week 8 | 31.67 [19.90 to 43.44] | 25.00 [14.04 to 35.96] | 18.75 [0.00 to 37.87] | 13.33 [0.00 to 30.54] | 11.76 [0.93 to 22.59] | 15.15 [2.92 to 27.38]
  Week 12 | 43.33 [30.79 to 55.87] | 31.67 [19.90 to 43.44] | 31.25 [8.54 to 53.96] | 20.00 [0.00 to 40.24] | 23.53 [9.27 to 37.79] | 12.12 [0.99 to 23.26]
  Week 16: number analyzed (Participants) | 59 | 60 | 16 | 15 | 34 | 33
  Week 16 | 44.07 [31.40 to 56.74] | 48.33 [35.69 to 60.98] | 31.25 [8.54 to 53.96] | 33.33 [9.48 to 57.19] | 14.71 [2.80 to 26.61] | 6.06 [0.00 to 14.20]
  Week 20 | 61.67 [49.36 to 73.97] | 53.33 [40.71 to 65.96] | 37.50 [13.78 to 61.22] | 40.00 [15.21 to 64.79] | 44.12 [27.43 to 60.81] | 45.45 [28.47 to 62.44]
  Week 28 | 56.67 [44.13 to 69.21] | 51.67 [39.02 to 64.31] | 43.75 [19.44 to 68.06] | 53.33 [28.09 to 78.58] | 41.18 [24.63 to 57.72] | 66.67 [50.58 to 82.75]
  Week 36 | 53.33 [40.71 to 65.96] | 56.67 [44.13 to 69.21] | 50.00 [25.50 to 74.50] | 66.67 [42.81 to 90.52] | 50.00 [33.19 to 66.81] | 57.58 [40.71 to 74.44]
  Week 44 | 56.67 [44.13 to 69.21] | 55.00 [42.41 to 67.59] | 43.75 [19.44 to 68.06] | 60.00 [35.21 to 84.79] | 58.82 [42.28 to 75.37] | 63.64 [47.22 to 80.05]
  Week 52 | 46.67 [34.04 to 59.29] | 58.33 [45.86 to 70.81] | 43.75 [19.44 to 68.06] | 46.67 [21.42 to 71.91] | 41.18 [24.63 to 57.72] | 51.52 [34.46 to 68.57]

5. Secondary Outcome: Percentage of Participants Achieving an ACR70 Response at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The American College of Rheumatology's definition for calculating improvement in rheumatoid arthritis (ACR70) was calculated as a ≥70% improvement in tender and swollen joint counts and ≥70% improvement in 3 of the 5 remaining ACR core set measures: patient pain assessment (a horizontal visual analog scale assessment of the patient's level of pain), patient global assessment (the patient's overall assessment of how the arthritis was doing by a visual analog scale), physician global assessment (a horizontal visual analog scale measure of the physician's assessment of the patient's current disease activity), patient self-assessed disability (a validated and reliable patient self-assessment instrument which measured physical functions in rheumatoid arthritis patients) and an acute-phase reactant (C-reactive protein level).
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: All participants who received at least 1 dose of the randomized study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Percentage of participants
  Week 2 | 3.33 [0.00 to 7.88] | 1.67 [0.00 to 4.91] | 2.94 [0.00 to 10.97] | 3.13 [0.00 to 11.65] | 1.43 [0.00 to 5.36] | 1.47 [0.00 to 5.52]
  Week 4 | 5.00 [0.00 to 10.51] | 5.00 [0.00 to 10.51] | 2.94 [0.00 to 10.97] | 3.13 [0.00 to 11.65] | 1.43 [0.00 to 5.36] | 1.47 [0.00 to 5.52]
  Week 8 | 11.67 [3.54 to 19.79] | 11.67 [3.54 to 19.79] | 6.25 [0.00 to 18.11] | 3.13 [0.00 to 11.65] | 2.94 [0.00 to 8.62] | 3.03 [0.00 to 8.88]
  Week 12 | 21.67 [11.24 to 32.09] | 18.33 [8.54 to 28.12] | 6.25 [0.00 to 18.11] | 6.67 [0.00 to 19.29] | 1.43 [0.00 to 5.36] | 9.09 [0.00 to 18.90]
  Week 16: number analyzed (Participants) | 59 | 60 | 16 | 15 | 34 | 33
  Week 16 | 23.73 [12.87 to 34.58] | 26.67 [15.48 to 37.86] | 6.25 [0.00 to 18.11] | 13.33 [0.00 to 30.54] | 1.43 [0.00 to 5.36] | 1.47 [0.00 to 5.52]
  Week 20 | 35.00 [22.93 to 47.07] | 30.00 [18.40 to 41.60] | 12.50 [0.00 to 28.70] | 20.00 [0.00 to 40.24] | 23.53 [9.27 to 37.79] | 27.27 [12.08 to 42.47]
  Week 28 | 36.67 [24.47 to 48.86] | 38.33 [26.03 to 50.64] | 18.75 [0.00 to 37.87] | 26.67 [4.29 to 49.05] | 23.53 [9.27 to 37.79] | 42.42 [25.56 to 59.29]
  Week 36 | 40.00 [27.60 to 52.40] | 35.00 [22.93 to 47.07] | 37.50 [13.78 to 61.22] | 26.67 [4.29 to 49.05] | 35.29 [19.23 to 51.36] | 39.39 [22.72 to 56.07]
  Week 44 | 46.67 [34.04 to 59.29] | 45.00 [32.41 to 57.59] | 37.50 [13.78 to 61.22] | 40.00 [15.21 to 64.79] | 23.53 [9.27 to 37.79] | 51.52 [34.46 to 68.57]
  Week 52 | 38.33 [26.03 to 50.64] | 45.00 [32.41 to 57.59] | 31.25 [8.54 to 53.96] | 26.67 [4.29 to 49.05] | 35.29 [19.23 to 51.36] | 42.42 [25.56 to 59.29]

6. Secondary Outcome: Change From Baseline in Tender/Painful Joint Count at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The tender/painful joints were assessed by a blinded assessor to determine the number of joints that were considered tender/painful using the following scale: Present/Absent/Not Done/Not Applicable (used for artificial or missing joints). Artificial joints was not assessed. Injected joints was counted according to their pre-injection status for the remainder of the study. The assessment was based on 68 joints. The score range was 0 to 68, with a higher score indicating a greater degree of tenderness. A negative change from baseline represents improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: "Overall Number of Participants Analyzed" indicated the evaluable population and included all participants who were randomized to the study and received at least one dose of the randomized study treatment. "Number Analyzed" included participants available in the evaluable population at each specified visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Units on a scale
  Week 2: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 2 | -3.33 (5.23) | -2.7 (4.49) | -4.7 (6.37) | 0.0 (2.70) | -1.9 (3.27) | -2.1 (5.41)
  Week 4: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 4 | -6.3 (7.96) | -5.1 (5.43) | -5.6 (8.93) | -2.8 (4.49) | -3.4 (5.47) | -4.3 (8.25)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | -9.4 (7.69) | -6.8 (6.49) | -7.9 (7.89) | -4.4 (6.42) | -5.0 (6.46) | -4.6 (8.41)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | -9.8 (8.19) | -8.7 (7.27) | -11.3 (7.32) | -6.2 (8.43) | -6.5 (6.69) | -6.4 (9.40)
  Week 16: number analyzed (Participants) | 56 | 57 | 14 | 13 | 31 | 31
  Week 16 | -11.1 (8.01) | -10.1 (7.33) | -12.0 (8.80) | -10.4 (8.69) | -6.5 (5.78) | -6.5 (7.81)
  Week 20: number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 | -12.2 (8.20) | -10.2 (6.60) | -13.6 (9.65) | -11.2 (10.95) | -8.8 (5.94) | -10.2 (7.41)
  Week 28: number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 | -12.6 (8.38) | -10.4 (7.04) | -14.9 (9.99) | -13.5 (12.21) | -9.6 (6.39) | -11.4 (8.13)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | -12.5 (8.66) | -10.7 (7.00) | -16.2 (9.45) | -13.8 (11.89) | -10.4 (6.12) | -11.4 (8.82)
  Week 44: number analyzed (Participants) | 47 | 54 | 10 | 12 | 27 | 28
  Week 44 | -13.6 (8.54) | -11.6 (7.91) | -17.9 (10.07) | -12.6 (13.23) | -11.3 (6.47) | -12.5 (9.15)
  Week 52: number analyzed (Participants) | 43 | 52 | 10 | 12 | 24 | 26
  Week 52 | -13.6 (9.11) | -11.9 (7.69) | -18.9 (10.74) | -13.0 (12.25) | -10.8 (5.53) | -12.2 (9.81)

7. Secondary Outcome: Change From Baseline in Swollen Joint Count at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The swollen joints were assessed by a blinded assessor to determine the number of joints that were considered swollen using the following scale: Present/Absent/Not Done/Not Applicable (used for artificial or missing joints). Artificial joints was not assessed. Injected joints was counted according to their pre-injection status for the remainder of the study. The assessment was based on 66 joints. The score range was 0 to 66, with a higher score indicating a greater degree of swelling. A negative change from baseline represents improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Units on a scale
  Week 2: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 2 | -2.3 (3.48) | -2.7 (3.73) | -4.6 (5.46) | -2.1 (3.31) | -2.0 (3.82) | -2.0 (3.95)
  Week 4: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 4 | -4.8 (4.42) | -4.3 (3.64) | -5.5 (5.51) | -5.2 (8.14) | -2.5 (3.11) | -3.6 (5.61)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | -6.5 (5.42) | -5.9 (4.50) | -7.9 (4.72) | -7.5 (7.54) | -4.4 (5.42) | -4.4 (5.95)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | -7.1 (5.89) | -6.7 (4.69) | -8.7 (6.97) | -8.7 (8.04) | -5.4 (5.26) | -4.7 (6.05)
  Week 16: number analyzed (Participants) | 56 | 57 | 14 | 13 | 31 | 31
  Week 16 | -8.0 (5.53) | -7.6 (5.10) | -8.9 (7.94) | -9.9 (8.98) | -6.7 (5.80) | -5.5 (6.74)
  Week 20: number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 | -8.5 (5.31) | -8.3 (5.12) | -10.5 (8.42) | -10.8 (9.10) | -8.0 (6.29) | -7.6 (5.15)
  Week 28: number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 | -8.2 (4.34) | -7.7 (5.27) | -10.0 (7.66) | -10.9 (9.00) | -7.2 (5.79) | -8.5 (5.83)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | -8.1 (4.35) | -8.1 (4.97) | -10.5 (7.55) | -11.1 (9.30) | -8.4 (5.60) | -8.9 (5.71)
  Week 44: number analyzed (Participants) | 47 | 54 | 10 | 12 | 27 | 28
  Week 44 | -8.3 (4.87) | -8.2 (5.05) | -10.5 (6.84) | -10.8 (9.93) | -8.3 (5.57) | -9.5 (5.51)
  Week 52: number analyzed (Participants) | 43 | 52 | 10 | 12 | 24 | 26
  Week 52 | -8.2 (4.84) | -8.1 (4.84) | -11.1 (7.68) | -10.7 (9.55) | -8.5 (5.76) | -9.2 (6.19)

8. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: Participants assessed the severity of their arthritis pain using a 100 millimeter (mm) visual analog scale (VAS) by placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponded to the magnitude of their pain. VAS data was rescaled prior to any calculation and analysis. Rescaled VAS score (mm) = (100 mm) × (length at mark in mm/overall length of line in mm). The score range was 0 mm to 100 mm, with a higher score indicating a higher degree of pain. A negative change from baseline represents improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
mm
  Week 2: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 2 | -7.6 (19.13) | -8.0 (17.96) | -5.3 (12.87) | 1.7 (21.20) | -2.3 (11.89) | -9.0 (17.52)
  Week 4: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 4 | -13.4 (23.39) | -18.5 (20.32) | -12.4 (22.60) | -7.9 (22.69) | -10.1 (18.67) | -9.6 (18.15)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | -20.6 (23.55) | -21.0 (22.46) | -14.3 (27.34) | -10.7 (25.94) | -16.9 (22.67) | -13.1 (22.88)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | -24.7 (25.72) | -22.8 (22.19) | -21.8 (24.25) | -14.9 (24.90) | -14.2 (24.54) | -12.3 (24.44)
  Week 16: number analyzed (Participants) | 57 | 57 | 14 | 13 | 31 | 31
  Week 16 | -28.4 (24.13) | -25.0 (22.58) | -26.5 (23.41) | -30.2 (20.55) | -13.7 (22.14) | -14.6 (20.16)
  Week 20: number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 | -29.5 (24.12) | -30.9 (22.91) | -29.3 (24.07) | -25.5 (29.91) | -32.1 (22.84) | -27.7 (26.78)
  Week 28: number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 | -29.7 (22.88) | -32.2 (25.21) | -34.6 (21.85) | -35.2 (24.79) | -29.6 (27.49) | -37.4 (25.54)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | -31.6 (25.14) | -31.3 (26.58) | -37.0 (29.87) | -33.5 (36.99) | -32.4 (21.11) | -38.5 (26.34)
  Week 44: number analyzed (Participants) | 47 | 54 | 10 | 12 | 27 | 28
  Week 44 | -32.8 (26.90) | -36.5 (26.87) | -41.6 (16.12) | -34.1 (39.69) | -35.0 (23.36) | -40.0 (26.21)
  Week 52: number analyzed (Participants) | 43 | 52 | 10 | 12 | 24 | 26
  Week 52 | -31.4 (26.39) | -35.5 (27.76) | -39.6 (21.95) | -34.9 (31.79) | -38.3 (22.84) | -38.5 (25.29)

9. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Arthritis at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: Participants answered the following question, "Considering all the ways your arthritis affects you, how are you feeling today?". The participant's response was recorded using a 100 mm visual analog scale (VAS) by placing a mark on the scale between 0 (very well) and 100 (very poorly). VAS data was rescaled prior to any calculation and analysis. Rescaled VAS score (mm) = (100 mm) × (length at mark in mm/overall length of line in mm). The score range was 0 mm to 100 mm, and a negative change from baseline represents improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
mm
  Week 2: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 2 | -6.3 (21.52) | -10.9 (17.85) | -5.4 (17.59) | 2.6 (19.66) | -0.1 (17.33) | -7.8 (17.02)
  Week 4: number analyzed (Participants) | 58 | 58 | 16 | 15 | 33 | 33
  Week 4 | -14.4 (25.55) | -20.5 (20.60) | -12.3 (18.09) | -8.9 (16.46) | -2.0 (20.76) | -3.3 (17.34)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | -19.4 (24.61) | -21.9 (24.29) | -14.0 (21.37) | -12.7 (19.88) | -11.0 (26.22) | -7.0 (22.38)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | -21.8 (26.15) | -26.2 (21.18) | -20.0 (24.36) | -12.4 (21.29) | -12.2 (26.00) | -8.0 (25.46)
  Week 16: number analyzed (Participants) | 57 | 57 | 14 | 13 | 31 | 31
  Week 16 | -27.8 (22.31) | -27.3 (21.62) | -26.1 (25.26) | -26.7 (19.05) | -9.3 (23.48) | -9.4 (21.11)
  Week 20: number analyzed (Participants) | 54 | 56 | 13 | 13 | 31 | 31
  Week 20 | -26.8 (23.84) | -31.4 (21.81) | -27.6 (23.49) | -22.8 (31.26) | -28.8 (25.44) | -25.5 (24.96)
  Week 28: number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 | -29.4 (20.78) | -34.0 (23.87) | -33.9 (22.09) | -33.7 (23.46) | -31.7 (24.10) | -33.9 (23.79)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | -30.1 (23.65) | -34.1 (26.03) | -37.2 (29.10) | -30.7 (39.29) | -28.5 (21.25) | -34.9 (24.80)
  Week 44: number analyzed (Participants) | 47 | 54 | 10 | 12 | 27 | 28
  Week 44 | -31.5 (24.77) | -34.9 (24.41) | -38.2 (22.88) | -33.0 (39.17) | -28.7 (23.22) | -35.6 (26.55)
  Week 52: number analyzed (Participants) | 43 | 52 | 10 | 12 | 24 | 26
  Week 52 | -32.0 (24.63) | -35.2 (28.60) | -36.8 (23.09) | -29.6 (32.56) | -34.9 (25.24) | -32.1 (28.85)

10. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritis at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The blinded assessor assessed the participant's overall arthritis appears at the time of each visit. This was an evaluation based on the participant's disease signs, functional capacity and physical examination, and was independent of the Patient's Global Assessment of Arthritis. The investigator's response was recorded using a 100 mm visual analog scale (VAS) by placing a mark on the scale between 0 (very good) and 100 (very poor). VAS data was rescaled prior to any calculation and analysis. Rescaled VAS score (mm) = (100 mm) × (length at mark in mm/overall length of line in mm). The score range was 0 mm to 100 mm, and a negative change from baseline represents improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
mm
  Week 2: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 2 | -9.2 (15.59) | -9.0 (14.87) | -9.9 (14.55) | -1.9 (10.79) | -3.4 (11.92) | -7.2 (13.64)
  Week 4: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 4 | -19.8 (18.98) | -17.6 (18.37) | -18.3 (22.31) | -11.1 (13.99) | -8.8 (17.67) | -9.5 (18.08)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | -30.6 (19.43) | -25.0 (18.02) | -28.7 (15.73) | -16.4 (21.08) | -16.3 (20.97) | -11.9 (17.94)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | -35.2 (19.92) | -30.1 (16.85) | -31.1 (20.62) | -21.2 (22.01) | -16.5 (21.57) | -13.7 (22.30)
  Week 16: number analyzed (Participants) | 56 | 57 | 14 | 13 | 31 | 31
  Week 16 | -37.7 (20.59) | -33.7 (17.89) | -31.2 (20.00) | -32.5 (23.98) | -16.5 (23.34) | -14.4 (27.76)
  Week 20: number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 | -41.8 (19.91) | -37.8 (19.48) | -38.7 (24.67) | -34.7 (26.16) | -31.0 (22.29) | -27.1 (25.41)
  Week 28: number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 | -42.0 (21.42) | -36.7 (21.91) | -47.6 (21.44) | -42.4 (23.28) | -32.7 (22.03) | -38.8 (20.53)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | -42.7 (22.92) | -36.8 (23.05) | -46.3 (22.42) | -43.4 (20.30) | -38.0 (19.52) | -42.6 (20.41)
  Week 44: number analyzed (Participants) | 47 | 54 | 10 | 12 | 27 | 28
  Week 44 | -44.5 (20.15) | -40.6 (22.19) | -51.9 (15.81) | -43.2 (25.55) | -36.4 (20.54) | -44.9 (20.40)
  Week 52: number analyzed (Participants) | 43 | 52 | 10 | 12 | 24 | 26
  Week 52 | -46.6 (21.73) | -43.4 (20.36) | -54.1 (15.18) | -42.7 (23.34) | -36.3 (21.01) | -41.9 (22.66)

11. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Disability Index (DI) at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The HAQ-DI assessed the degree of difficulty a participant experienced in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2-3 items. For each question in the questionnaire, the level of difficulty is scored from 0 to 3 with 0 representing "no difficulty," 1 as "some difficulty," 2 as "much difficulty," and 3 as "unable to do". Any activity that requires assistance from another individual or requires the use of an assistive device adjusts to a minimum score of 2 to represent a more limited functional status. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range was 0 to 3, with a higher score indicating more difficulty in performing daily living activities. A negative change from baseline represents improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Units on a scale
  Week 2: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 2 | -0.133 (0.4273) | -0.177 (0.3489) | -0.195 (0.2886) | -0.117 (0.4212) | -0.030 (0.4572) | -0.170 (0.3091)
  Week 4: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 4 | -0.248 (0.5341) | -0.315 (0.3777) | -0.180 (0.2090) | -0.217 (0.3356) | -0.095 (0.4931) | -0.170 (0.3305)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | -0.343 (0.5690) | -0.421 (0.4103) | -0.188 (0.4472) | -0.277 (0.3609) | -0.184 (0.4959) | -0.249 (0.4465)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | -0.366 (0.5701) | -0.478 (0.4167) | -0.214 (0.4230) | -0.304 (0.2930) | -0.121 (0.4910) | -0.239 (0.4660)
  Week 16: number analyzed (Participants) | 57 | 57 | 14 | 13 | 31 | 31
  Week 16 | -0.474 (0.5158) | -0.509 (0.3994) | -0.321 (0.3914) | -0.375 (0.3385) | -0.109 (0.5271) | -0.246 (0.3729)
  Week 20: number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 | -0.466 (0.5546) | -0.576 (0.4906) | -0.404 (0.4681) | -0.308 (0.4610) | -0.363 (0.4983) | -0.472 (0.4934)
  Week 28: number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 | -0.524 (0.5412) | -0.583 (0.5262) | -0.519 (0.4531) | -0.490 (0.5064) | -0.422 (0.4811) | -0.517 (0.5520)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | -0.520 (0.6051) | -0.594 (0.4990) | -0.577 (0.5740) | -0.519 (0.5633) | -0.329 (0.3816) | -0.547 (0.5867)
  Week 44: number analyzed (Participants) | 47 | 54 | 10 | 12 | 27 | 28
  Week 44 | -0.521 (0.6197) | -0.581 (0.5321) | -0.563 (0.3830) | -0.510 (0.5576) | -0.370 (0.4210) | -0.576 (0.5757)
  Week 52: number analyzed (Participants) | 43 | 52 | 10 | 12 | 24 | 26
  Week 52 | -0.503 (0.6023) | -0.567 (0.4866) | -0.500 (0.5137) | -0.552 (0.5041) | -0.411 (0.3695) | -0.514 (0.5704)

12. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein (hsCRP) at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: C-reactive protein (hsCRP) is an acute phase reactant, which is indicative of inflammation and of its severity. Blood samples were obtained at Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52 for determination of hsCRP.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: "Overall Number of Participants Analyzed" included all the participants in the pharmacodynamic (PD) analysis population who received at least one dose of randomized study treatment and in whom at least one value of the PD parameter of interest was reported. "Number Analyzed" included participants available in the PD analysis population at each specified visit.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
milligram per liter (mg/L)
  Week 2: number analyzed (Participants) | 58 | 58 | 16 | 15 | 33 | 33
  Week 2 | -4.420 (8.9409) | -3.696 (11.9628) | -6.023 (19.1126) | -0.595 (1.4661) | -1.641 (10.4224) | 1.462 (7.8966)
  Week 4: number analyzed (Participants) | 59 | 57 | 16 | 15 | 33 | 33
  Week 4 | -3.645 (11.8144) | -5.543 (11.9617) | -6.134 (19.5633) | -1.324 (1.9735) | 0.010 (7.0206) | 1.206 (5.4423)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | -3.828 (10.8093) | -5.102 (11.5408) | -6.029 (19.9534) | -0.573 (2.6595) | -2.598 (10.7270) | 0.927 (6.2062)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | -3.759 (11.0481) | -5.881 (12.9484) | -7.335 (22.0149) | -1.177 (3.4854) | -1.061 (11.1944) | 1.021 (6.6025)
  Week 16: number analyzed (Participants) | 56 | 57 | 14 | 13 | 30 | 31
  Week 16 | -3.695 (8.1064) | -5.809 (13.6463) | -5.420 (21.9622) | 1.060 (8.7842) | -2.218 (11.6164) | -0.762 (6.5779)
  Week 20: number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 | -4.581 (10.5026) | -6.014 (14.7723) | -7.879 (24.2763) | -0.989 (3.6969) | -5.982 (10.4711) | -4.718 (7.1896)
  Week 28: number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 | -4.277 (12.9069) | -6.362 (13.6372) | -8.679 (24.9759) | -1.300 (3.7971) | -6.112 (10.6756) | -5.484 (10.0475)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | -4.899 (10.3015) | -5.940 (14.4219) | -9.461 (25.7767) | -1.814 (3.0658) | -6.247 (9.8145) | -5.029 (9.1947)
  Week 44: number analyzed (Participants) | 46 | 54 | 10 | 12 | 27 | 28
  Week 44 | -5.543 (11.7058) | -6.215 (14.2493) | -2.196 (2.2859) | -0.987 (3.7325) | -4.690 (9.9495) | -0.711 (13.7530)
  Week 52: number analyzed (Participants) | 41 | 50 | 10 | 12 | 23 | 26
  Week 52 | -5.167 (13.3963) | -4.880 (14.1148) | -1.586 (3.0576) | -2.028 (3.2177) | -4.324 (7.7335) | -4.722 (9.3318)

13. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index 75 (PASI 75) Response at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percentage of body surface area (BSA) affected. Assessments of lesion Severity Score and Area Score are performed separately for each of the four body regions: head (including neck), upper limbs, trunk (including axillae and groin), and lower limbs (including buttocks). In each body region, the sum of the lesion Severity Scores for erythema, induration and scaling is multiplied by the Area Score which represents the percentage of this area involved by psoriasis, multiplied by a weighting factor (head 0.1; upper limbs 0.2; trunk 0.3; lower limbs 0.4). The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 75 indicates a 75% or greater reduction in PASI scores from baseline.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: "Overall Number of Participants Analyzed" included a subgroup of participants in the evaluable population (participants who were randomized to the study and received at least one dose of the randomized study treatment) with baseline BSA ≥3% and PASI >0 . "Number Analyzed" included participants available in the evaluable population at each specified visit with baseline BSA ≥3% and PASI >0.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 40 | 39 | 12 | 9 | 22 | 19
Percentage of participants
  Week 2 | 5.00 [0.00 to 11.75] | 2.56 [0.00 to 7.52] | 3.85 [0.00 to 14.30] | 11.11 [0.00 to 31.64] | 2.17 [0.00 to 8.13] | 5.26 [0.00 to 15.30]
  Week 4 | 30.00 [15.80 to 44.20] | 12.82 [2.33 to 23.31] | 3.85 [0.00 to 14.30] | 11.11 [0.00 to 31.64] | 4.55 [0.00 to 13.25] | 5.26 [0.00 to 15.30]
  Week 8 | 45.00 [29.58 to 60.42] | 41.03 [25.59 to 56.46] | 25.00 [0.50 to 49.50] | 11.11 [0.00 to 31.64] | 9.09 [0.00 to 21.10] | 15.79 [0.00 to 32.19]
  Week 12 | 60.00 [44.82 to 75.18] | 48.72 [33.03 to 64.41] | 33.33 [6.66 to 60.01] | 33.33 [2.54 to 64.13] | 18.18 [2.06 to 34.30] | 21.05 [2.72 to 39.38]
  Week 16: number analyzed (Participants) | 39 | 39 | 12 | 9 | 22 | 19
  Week 16 | 69.23 [54.75 to 83.72] | 58.97 [43.54 to 74.41] | 58.33 [30.44 to 86.23] | 55.56 [23.09 to 88.02] | 22.73 [5.22 to 40.24] | 26.32 [6.52 to 46.12]
  Week 20 | 72.50 [58.66 to 86.34] | 61.54 [46.27 to 76.81] | 66.67 [39.99 to 93.34] | 55.56 [23.09 to 88.02] | 54.55 [33.74 to 75.35] | 36.84 [15.15 to 58.53]
  Week 28 | 70.00 [55.80 to 84.20] | 51.28 [35.59 to 66.97] | 91.67 [76.03 to 100.00] | 77.78 [50.62 to 100.00] | 63.64 [43.54 to 83.74] | 63.16 [41.47 to 84.85]
  Week 36 | 70.00 [55.80 to 84.20] | 64.10 [49.05 to 79.16] | 96.15 [85.70 to 100.00] | 88.89 [68.36 to 100.00] | 59.09 [38.55 to 79.64] | 47.37 [24.92 to 69.82]
  Week 44 | 75.00 [61.58 to 88.42] | 66.67 [51.87 to 81.46] | 75.00 [50.50 to 99.50] | 55.56 [23.09 to 88.02] | 63.64 [43.54 to 83.74] | 63.16 [41.47 to 84.85]
  Week 52 | 65.00 [50.22 to 79.78] | 66.67 [51.87 to 81.46] | 66.67 [39.99 to 93.34] | 66.67 [35.87 to 97.46] | 50.00 [29.11 to 70.89] | 57.89 [35.69 to 80.10]

14. Secondary Outcome: Percentage of Participants Achieving a PASI 90 Response at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percentage of body surface area (BSA) affected. Assessments of lesion Severity Score and Area Score are performed separately for each of the four body regions: head (including neck), upper limbs, trunk (including axillae and groin), and lower limbs (including buttocks). In each body region, the sum of the lesion Severity Scores for erythema, induration and scaling is multiplied by the Area Score which represents the percentage of this area involved by psoriasis, multiplied by a weighting factor (head 0.1; upper limbs 0.2; trunk 0.3; lower limbs 0.4). The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 90 indicates a 90% or greater reduction in PASI scores from baseline.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 40 | 39 | 12 | 9 | 22 | 19
Percentage of participants
  Week 2 | 1.22 [0.00 to 4.58] | 1.25 [0.00 to 4.69] | 3.85 [0.00 to 14.30] | 11.11 [0.00 to 31.64] | 2.17 [0.00 to 8.13] | 2.50 [0.00 to 9.34]
  Week 4 | 17.50 [5.72 to 29.28] | 5.13 [0.00 to 12.05] | 3.85 [0.00 to 14.30] | 11.11 [0.00 to 31.64] | 4.55 [0.00 to 13.25] | 2.50 [0.00 to 9.34]
  Week 8 | 35.00 [20.22 to 49.78] | 17.95 [5.90 to 29.99] | 16.67 [0.00 to 37.75] | 11.11 [0.00 to 31.64] | 2.17 [0.00 to 8.13] | 5.26 [0.00 to 15.30]
  Week 12 | 47.50 [32.02 to 62.98] | 25.64 [11.94 to 39.35] | 16.67 [0.00 to 37.75] | 22.22 [0.00 to 49.38] | 2.17 [0.00 to 8.13] | 10.53 [0.00 to 24.33]
  Week 16: number analyzed (Participants) | 39 | 39 | 12 | 9 | 22 | 19
  Week 16 | 53.85 [38.20 to 69.49] | 33.33 [18.54 to 48.13] | 33.33 [6.66 to 60.01] | 33.33 [2.54 to 64.13] | 9.09 [0.00 to 21.10] | 15.79 [0.00 to 32.19]
  Week 20 | 50.00 [34.51 to 65.49] | 43.59 [28.03 to 59.15] | 50.00 [21.71 to 78.29] | 44.44 [11.98 to 76.91] | 18.18 [2.06 to 34.30] | 26.32 [6.52 to 46.12]
  Week 28 | 52.50 [37.02 to 67.98] | 38.46 [23.19 to 53.73] | 58.33 [30.44 to 86.23] | 44.44 [11.98 to 76.91] | 50.00 [29.11 to 70.89] | 31.58 [10.68 to 52.48]
  Week 36 | 62.50 [47.50 to 77.50] | 48.72 [33.03 to 64.41] | 83.33 [62.25 to 100.00] | 66.67 [35.87 to 97.46] | 45.45 [24.65 to 66.26] | 36.84 [15.15 to 58.53]
  Week 44 | 52.50 [37.02 to 67.98] | 48.72 [33.03 to 64.41] | 66.67 [39.99 to 93.34] | 44.44 [11.98 to 76.91] | 50.00 [29.11 to 70.89] | 52.63 [30.18 to 75.08]
  Week 52 | 40.00 [24.82 to 55.18] | 56.41 [40.85 to 71.97] | 66.67 [39.99 to 93.34] | 55.56 [23.09 to 88.02] | 45.45 [24.65 to 66.26] | 47.37 [24.92 to 69.82]

15. Secondary Outcome: Percentage of Participants Achieving a PASI 100 Response at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percentage of body surface area (BSA) affected. Assessments of lesion Severity Score and Area Score are performed separately for each of the four body regions: head (including neck), upper limbs, trunk (including axillae and groin), and lower limbs (including buttocks). In each body region, the sum of the lesion Severity Scores for erythema, induration and scaling is multiplied by the Area Score which represents the percentage of this area involved by psoriasis, multiplied by a weighting factor (head 0.1; upper limbs 0.2; trunk 0.3; lower limbs 0.4). The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI 100 indicates a 100% reduction in PASI scores from baseline.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 40 | 39 | 12 | 9 | 22 | 19
Percentage of participants
  Week 2 | 1.22 [0.00 to 4.58] | 1.25 [0.00 to 4.69] | 3.85 [0.00 to 14.30] | 11.11 [0.00 to 31.64] | 2.17 [0.00 to 8.13] | 2.50 [0.00 to 9.34]
  Week 4 | 7.50 [0.00 to 15.66] | 1.25 [0.00 to 4.69] | 3.85 [0.00 to 14.30] | 5.00 [0.00 to 18.51] | 4.55 [0.00 to 13.25] | 2.50 [0.00 to 9.34]
  Week 8 | 20.00 [7.60 to 32.40] | 5.13 [0.00 to 12.05] | 8.33 [0.00 to 23.97] | 11.11 [0.00 to 31.64] | 2.17 [0.00 to 8.13] | 2.50 [0.00 to 9.34]
  Week 12 | 35.00 [20.22 to 49.78] | 7.69 [0.00 to 16.06] | 8.33 [0.00 to 23.97] | 11.11 [0.00 to 31.64] | 2.17 [0.00 to 8.13] | 5.26 [0.00 to 15.30]
  Week 16: number analyzed (Participants) | 39 | 39 | 12 | 9 | 22 | 19
  Week 16 | 35.90 [20.84 to 50.95] | 15.38 [4.06 to 26.71] | 16.67 [0.00 to 37.75] | 33.33 [2.54 to 64.13] | 9.09 [0.00 to 21.10] | 10.53 [0.00 to 24.33]
  Week 20 | 27.50 [13.66 to 41.34] | 35.90 [20.84 to 50.95] | 33.33 [6.66 to 60.01] | 44.44 [11.98 to 76.91] | 13.64 [0.00 to 27.98] | 10.53 [0.00 to 24.33]
  Week 28 | 35.00 [20.22 to 49.78] | 30.77 [16.28 to 45.25] | 50.00 [21.71 to 78.29] | 44.44 [11.98 to 76.91] | 40.91 [20.36 to 61.45] | 21.05 [2.72 to 39.38]
  Week 36 | 40.00 [24.82 to 55.18] | 35.90 [20.84 to 50.95] | 50.00 [21.71 to 78.29] | 55.56 [23.09 to 88.02] | 36.36 [16.26 to 56.46] | 21.05 [2.72 to 39.38]
  Week 44 | 30.00 [15.80 to 44.20] | 41.03 [25.59 to 56.46] | 58.33 [30.44 to 86.23] | 44.44 [11.98 to 76.91] | 31.82 [12.36 to 51.28] | 42.11 [19.90 to 64.31]
  Week 52 | 35.00 [20.22 to 49.78] | 38.46 [23.19 to 53.73] | 41.67 [13.77 to 69.56] | 33.33 [2.54 to 64.13] | 36.36 [16.26 to 56.46] | 42.11 [19.90 to 64.31]

16. Secondary Outcome: Change From Baseline in the Enthesitis Score (Using the Spondyloarthritis Research Consortium of Canada [SPARCC] Enthesitis Index) at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The SPARCC Enthesitis Index examines tenderness at sixteen sites: medial epicondyle humerus, lateral epicondyle humerus, supraspinatus insertion into greater tuberosity of humerus, greater trochanter, quadriceps insertion into superior border of patella, patellar ligament insertion into inferior pole of patella or tibial tubercle (considered 1 site for scoring purposes), Achilles tendon insertion into calcaneum and plantar fascia insertion into calcaneum. Each site is classified on a dichotomous basis as either tender (score=1) or not tender (score=0). The SPARCC Enthesitis Index scores range from 0-16, with higher scores indicating higher disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: "Overall Number of Participants Analyzed" included all the participants in the evaluable population (participants who were randomized to the study and received at least one dose of the randomized study treatment) with baseline SPARCC enthesitis score>0. "Number Analyzed" included participants available in the evaluable population at each specified treatment timepoints with baseline SPARCC enthesitis score >0.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 38 | 34 | 11 | 9 | 21 | 19
Units on a scale
  Week 2: number analyzed (Participants) | 37 | 32 | 11 | 9 | 20 | 19
  Week 2 | -0.6 (1.55) | -0.3 (2.73) | -1.4 (1.86) | 0.0 (1.12) | -0.2 (1.79) | -0.3 (2.67)
  Week 4: number analyzed (Participants) | 37 | 32 | 11 | 9 | 20 | 19
  Week 4 | -1.4 (2.41) | -0.9 (2.32) | -1.3 (2.37) | 0.0 (1.41) | -1.0 (2.29) | -1.0 (2.81)
  Week 8: number analyzed (Participants) | 36 | 31 | 11 | 8 | 19 | 19
  Week 8 | -1.9 (2.11) | -1.9 (2.23) | -1.4 (1.80) | -1.0 (1.07) | -1.1 (2.50) | -1.2 (2.53)
  Week 12: number analyzed (Participants) | 37 | 31 | 9 | 8 | 18 | 19
  Week 12 | -2.1 (2.49) | -1.6 (2.22) | -2.7 (1.73) | -1.3 (1.04) | -1.7 (2.52) | -1.1 (3.00)
  Week 16: number analyzed (Participants) | 36 | 31 | 9 | 8 | 18 | 18
  Week 16 | -2.1 (2.68) | -1.3 (1.89) | -3.1 (1.27) | -0.3 (2.71) | -1.8 (2.94) | -1.2 (2.79)
  Week 20: number analyzed (Participants) | 36 | 31 | 9 | 8 | 18 | 18
  Week 20 | -2.3 (2.66) | -1.9 (2.29) | -3.2 (3.03) | -1.3 (0.89) | -2.1 (2.24) | -1.9 (2.71)
  Week 28: number analyzed (Participants) | 33 | 31 | 9 | 8 | 16 | 18
  Week 28 | -2.4 (2.68) | -2.3 (2.60) | -3.8 (2.05) | -1.4 (1.19) | -2.5 (2.97) | -3.1 (2.60)
  Week 36: number analyzed (Participants) | 31 | 31 | 9 | 8 | 14 | 18
  Week 36 | -2.6 (2.70) | -2.3 (2.28) | -3.8 (2.79) | -1.6 (1.06) | -2.1 (2.51) | -2.8 (2.60)
  Week 44: number analyzed (Participants) | 29 | 31 | 8 | 8 | 14 | 17
  Week 44 | -2.9 (2.56) | -2.4 (2.53) | -3.3 (1.67) | -1.6 (1.06) | -2.1 (2.57) | -3.2 (2.44)
  Week 52: number analyzed (Participants) | 27 | 30 | 8 | 8 | 13 | 15
  Week 52 | -3.1 (2.55) | -2.4 (2.34) | -4.8 (2.76) | -1.5 (0.76) | -2.2 (1.74) | -3.6 (2.59)

17. Secondary Outcome: Change From Baseline in the Enthesitis Score (Using the Leeds Enthesitis Index) at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The Leeds Enthesitis Index (LEI) examines tenderness at six sites: lateral epicondyle humerus, medial femoral condyle and Achilles tendon insertion. Each site is assessed as either tender (score=1) or not tender (score=0). The LEI scores range from 0-6, with higher scores indicating higher disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: "Overall Number of Participants Analyzed" included all the participants in the evaluable population (participants who were randomized to the study and received at least one dose of the randomized study treatment) with baseline leeds enthesitis score>0. "Number Analyzed" included participants available in the evaluable population at each specified treatment timepoints with baseline leeds enthesitis score>0.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 29 | 28 | 10 | 8 | 20 | 15
Units on a scale
  Week 2: number analyzed (Participants) | 28 | 26 | 10 | 8 | 20 | 15
  Week 2 | -0.4 (0.95) | -0.4 (1.53) | -0.5 (1.27) | 0.0 (0.53) | -0.1 (1.12) | -0.3 (0.82)
  Week 4: number analyzed (Participants) | 28 | 26 | 10 | 8 | 20 | 15
  Week 4 | -0.7 (1.56) | -0.9 (1.48) | -1.0 (1.25) | -0.1 (0.99) | -0.4 (0.75) | -0.9 (1.62)
  Week 8: number analyzed (Participants) | 27 | 25 | 10 | 7 | 19 | 15
  Week 8 | -1.3 (1.43) | -1.2 (1.47) | -0.5 (1.78) | -0.4 (0.98) | -0.5 (1.31) | -0.7 (1.49)
  Week 12: number analyzed (Participants) | 28 | 25 | 9 | 7 | 18 | 15
  Week 12 | -1.2 (1.93) | -1.5 (1.42) | -1.0 (1.22) | -1.1 (0.90) | -0.9 (0.94) | -0.9 (1.79)
  Week 16: number analyzed (Participants) | 27 | 25 | 9 | 7 | 18 | 14
  Week 16 | -1.4 (1.63) | -1.5 (1.45) | -1.2 (0.83) | -0.1 (2.12) | -0.9 (1.13) | -0.9 (1.54)
  Week 20: number analyzed (Participants) | 27 | 25 | 9 | 7 | 18 | 14
  Week 20 | -1.6 (1.52) | -1.3 (1.80) | -1.7 (2.65) | -0.9 (0.90) | -1.1 (0.90) | -1.4 (1.91)
  Week 28: number analyzed (Participants) | 25 | 25 | 9 | 7 | 16 | 14
  Week 28 | -1.4 (1.56) | -1.7 (1.57) | -1.9 (2.20) | -1.3 (0.76) | -1.1 (1.20) | -1.7 (1.54)
  Week 36: number analyzed (Participants) | 23 | 25 | 9 | 7 | 14 | 14
  Week 36 | -1.9 (1.36) | -1.8 (1.59) | -2.3 (1.50) | -1.1 (0.90) | -1.1 (1.17) | -1.7 (1.44)
  Week 44: number analyzed (Participants) | 22 | 25 | 8 | 7 | 14 | 14
  Week 44 | -1.8 (1.47) | -1.8 (1.65) | -2.3 (1.04) | -1.3 (0.76) | -1.2 (1.19) | -1.9 (1.41)
  Week 52: number analyzed (Participants) | 20 | 24 | 8 | 7 | 13 | 12
  Week 52 | -2.0 (1.54) | -1.7 (1.40) | -2.5 (0.93) | -1.0 (0.82) | -1.2 (0.73) | -1.8 (1.70)

18. Secondary Outcome: Change From Baseline in the Dactylitis Severity Score (DSS) at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The number of digits in hands and feet with dactylitis was evaluated by a blinded assessor. In addition, dactylitis severity was scored based upon digit tenderness using a scale of 0-3, where 0 = no tenderness to 3 = extreme tenderness, in each digit of the hands and feet. The range of total dactylitis scores was 0-60, with higher scores indicating greater severity. A negative change from baseline represents improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: "Overall Number of Participants Analyzed" included all the participants in evaluable population (participants who were randomized to the study and received at least one dose of the randomized study treatment) with baseline DSS >0. "Number Analyzed" included participants available in the evaluable population at each specified treatment timepoints with baseline DSS >0.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 14 | 19 | 3 | 6 | 12 | 19
Units on a scale
  Week 2: number analyzed (Participants) | 14 | 17 | 3 | 6 | 12 | 9
  Week 2 | -0.2 (2.36) | -0.7 (2.54) | -2.7 (4.62) | -0.5 (1.38) | -0.7 (1.61) | 0.2 (2.28)
  Week 4: number analyzed (Participants) | 14 | 17 | 3 | 6 | 12 | 9
  Week 4 | -1.6 (3.30) | -2.2 (3.15) | -3.3 (3.21) | -0.8 (1.17) | -1.2 (2.59) | -0.3 (3.12)
  Week 8: number analyzed (Participants) | 14 | 17 | 3 | 6 | 11 | 9
  Week 8 | -3.5 (4.31) | -4.0 (3.22) | -4.3 (4.16) | -1.7 (1.37) | -2.5 (6.14) | -1.8 (2.82)
  Week 12: number analyzed (Participants) | 14 | 17 | 3 | 6 | 10 | 9
  Week 12 | -4.4 (3.34) | -4.5 (3.30) | -4.3 (4.93) | -3.2 (3.43) | -4.8 (7.07) | -2.8 (4.49)
  Week 16: number analyzed (Participants) | 14 | 17 | 3 | 6 | 10 | 9
  Week 16 | -3.7 (3.85) | -4.9 (4.06) | -4.7 (6.35) | -3.7 (4.13) | -5.4 (7.44) | -2.9 (6.01)
  Week 20: number analyzed (Participants) | 13 | 17 | 3 | 6 | 10 | 9
  Week 20 | -4.4 (3.31) | -4.6 (4.23) | -5.3 (5.86) | -3.7 (4.13) | -7.0 (7.44) | -4.4 (6.11)
  Week 28: number analyzed (Participants) | 12 | 17 | 3 | 6 | 9 | 9
  Week 28 | -3.8 (3.67) | -5.1 (4.08) | -5.3 (5.86) | -3.7 (4.13) | -6.6 (7.18) | -4.7 (7.05)
  Week 36: number analyzed (Participants) | 10 | 17 | 3 | 6 | 9 | 8
  Week 36 | -4.2 (4.02) | -5.1 (4.26) | -5.7 (5.69) | -3.7 (4.13) | -6.8 (7.34) | -5.3 (7.40)
  Week 44: number analyzed (Participants) | 10 | 17 | 3 | 6 | 9 | 8
  Week 44 | -5.0 (3.65) | -5.4 (4.01) | -5.7 (5.69) | -3.7 (4.13) | -6.8 (7.34) | -5.3 (7.40)
  Week 52: number analyzed (Participants) | 10 | 17 | 3 | 6 | 8 | 6
  Week 52 | -5.0 (3.65) | -5.4 (4.05) | -5.7 (5.69) | -3.7 (4.13) | -5.0 (5.40) | -5.7 (8.62)

19. Secondary Outcome: Change From Baseline in the Nail Psoriasis Severity Index (NAPSI) Score at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: A target finger nail was evaluated by the blinded assessor using the NAPSI scale. At the baseline visit, the worst case fingernail was chosen and the same nail was evaluated consistently through the entire study. Each quadrant of the target nail was graded for nail matrix psoriasis (including any of the following parameters: pitting, leukonychia, red spots in lunula, nail plate crumbling) and nail bed psoriasis (including any of the following parameters: onycholysis, splinter hemorrhages, oil drop (salmon patch) discoloration, nail bed hyperkeratosis). The target nail NAPSI scores range from 0 to 8, with higher scores indicating higher disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: "Overall Number of Participants Analyzed" included all the participants in evaluable population (participants who were randomized to the study and received at least one dose of the randomized study treatment) with baseline NAPSI>0. "Number Analyzed" included participants available in the evaluable population at each specified treatment timepoints with baseline NAPSI>0.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 36 | 40 | 10 | 8 | 25 | 16
Units on a scale
  Week 2: number analyzed (Participants) | 36 | 38 | 10 | 8 | 23 | 16
  Week 2 | -0.4 (1.55) | 0.1 (0.65) | -0.4 (0.52) | 0.3 (0.71) | -0.2 (1.04) | 0.1 (0.25)
  Week 4: number analyzed (Participants) | 36 | 38 | 10 | 8 | 23 | 16
  Week 4 | -1.0 (2.09) | -0.5 (1.70) | -0.9 (1.10) | -0.3 (0.46) | -1.0 (2.16) | -0.3 (0.95)
  Week 8: number analyzed (Participants) | 35 | 38 | 10 | 7 | 22 | 16
  Week 8 | -2.0 (2.40) | -1.0 (1.49) | -1.1 (1.52) | -1.1 (1.57) | -1.3 (2.55) | -0.6 (1.55)
  Week 12: number analyzed (Participants) | 35 | 38 | 8 | 7 | 22 | 16
  Week 12 | -2.8 (2.54) | -1.8 (2.43) | -0.5 (2.88) | -1.9 (2.97) | -1.2 (2.62) | -1.3 (1.82)
  Week 16: number analyzed (Participants) | 34 | 38 | 8 | 7 | 22 | 15
  Week 16 | -3.2 (2.71) | -1.7 (2.54) | -1.5 (2.00) | -2.9 (3.08) | -1.4 (2.61) | -1.6 (1.76)
  Week 20: number analyzed (Participants) | 35 | 38 | 7 | 7 | 22 | 15
  Week 20 | -3.7 (2.82) | -2.3 (2.31) | -2.1 (2.41) | -3.1 (2.97) | -2.0 (2.61) | -1.9 (1.81)
  Week 28: number analyzed (Participants) | 32 | 38 | 7 | 7 | 20 | 14
  Week 28 | -3.9 (2.90) | -2.4 (2.56) | -3.1 (2.12) | -3.3 (2.93) | -2.2 (2.59) | -2.5 (1.83)
  Week 36: number analyzed (Participants) | 29 | 38 | 7 | 7 | 19 | 14
  Week 36 | -3.9 (3.06) | -2.5 (2.51) | -3.3 (1.98) | -3.3 (3.15) | -2.8 (2.71) | -2.9 (1.75)
  Week 44: number analyzed (Participants) | 28 | 37 | 5 | 6 | 19 | 13
  Week 44 | -4.2 (2.77) | -2.8 (2.47) | -4.2 (2.05) | -3.8 (3.19) | -2.8 (2.61) | -2.6 (1.71)
  Week 52: number analyzed (Participants) | 25 | 36 | 5 | 6 | 17 | 12
  Week 52 | -4.2 (2.62) | -2.6 (2.80) | -3.6 (2.07) | -3.7 (3.27) | -3.1 (2.91) | -2.7 (1.30)

20. Secondary Outcome: Change From Baseline in the Patient's Global Joint and Skin Assessment-Visual Analog Scale (PGJS-VAS) at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: Participant's perception of disease was assessed using a 100 mm visual analog scale (VAS) by placing a mark on the scale between 0 (excellent) and 100 (poor). The rating corresponded to the way in which the participant felt over the past week in terms of how they were affected by their: 1) psoriasis and arthritis (global, PGA); 2) arthritis only (PJA) and 3) psoriasis only (PSA). Rescaled VAS score was used. Rescaled VAS score (mm) = (100 mm) × (length at mark in mm/overall length of line in mm). A negative change from baseline represents improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
mm
  Week 2: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 2 | -8.9 (26.88) | -11.6 (22.31) | -4.9 (12.42) | -0.5 (12.41) | -3.3 (14.50) | -7.1 (17.44)
  Week 4: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 4 | -17.0 (24.83) | -18.8 (25.42) | -13.2 (18.69) | -7.1 (21.61) | -11.6 (22.07) | -6.2 (24.53)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | -21.1 (26.95) | -19.7 (27.56) | -12.0 (26.52) | -16.4 (25.36) | -16.8 (26.21) | -8.1 (24.41)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | -25.1 (28.18) | -25.3 (23.75) | -18.0 (21.42) | -17.6 (23.70) | -14.4 (28.78) | -9.5 (23.74)
  Week 16: number analyzed (Participants) | 57 | 57 | 14 | 13 | 31 | 31
  Week 16 | -29.0 (24.78) | -24.5 (25.43) | -23.9 (21.10) | -27.8 (21.23) | -11.7 (23.36) | -9.9 (23.87)
  Week 20: number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 | -29.1 (24.08) | -30.5 (23.29) | -27.3 (24.19) | -22.6 (27.92) | -36.3 (22.12) | -26.3 (29.72)
  Week 28: number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 | -30.0 (24.53) | -29.7 (28.36) | -37.2 (22.80) | -38.8 (25.73) | -37.3 (25.35) | -37.2 (24.64)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | -29.1 (27.81) | -29.6 (27.90) | -42.0 (26.37) | -33.7 (27.04) | -36.0 (22.02) | -39.4 (26.35)
  Week 44: number analyzed (Participants) | 47 | 54 | 10 | 12 | 27 | 28
  Week 44 | -33.6 (28.52) | -32.4 (28.81) | -41.9 (19.08) | -36.8 (30.62) | -38.2 (26.65) | -42.1 (27.08)
  Week 52: number analyzed (Participants) | 43 | 52 | 10 | 12 | 24 | 26
  Week 52 | -33.3 (28.68) | -32.7 (29.77) | -35.6 (26.94) | -33.9 (33.45) | -39.1 (23.78) | -38.3 (30.58)

21. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) at Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The FACIT-F Scale is a patient completed questionnaire consisting of 13 items that assess fatigue. Participants responded to each item on a 5-point scale based on their experience of fatigue during the past 7 days (0 = not at all; 1 = a little bit; 2 =somewhat; 3 = quite a bit; 4 = very much). Instrument scoring yielded a range from 0 to 52 (negatively worded items were reversed during analysis), with higher scores representing better participant status (less fatigue).
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Units on a scale
  Week 2: number analyzed (Participants) | 58 | 58 | 16 | 15 | 33 | 33
  Week 2 | 2.0 (5.82) | 3.1 (5.85) | 0.9 (2.60) | 1.2 (6.45) | 0.9 (6.95) | 2.7 (6.07)
  Week 4: number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 4 | 2.4 (7.47) | 5.7 (7.34) | 3.7 (5.40) | 3.7 (8.30) | 3.0 (10.76) | 2.5 (6.98)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | 4.2 (8.03) | 5.6 (8.44) | 3.6 (5.78) | 3.8 (6.24) | 3.2 (10.31) | 3.7 (9.92)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | 4.7 (10.17) | 7.3 (7.96) | 3.2 (4.10) | 6.1 (7.85) | 5.5 (9.55) | 3.8 (9.85)
  Week 16: number analyzed (Participants) | 57 | 57 | 14 | 13 | 31 | 31
  Week 16 | 5.6 (7.74) | 7.1 (9.41) | 4.4 (5.40) | 6.0 (6.89) | 4.7 (8.10) | 4.7 (8.99)
  Week 20: number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 | 6.6 (8.69) | 9.5 (8.20) | 7.2 (5.86) | 7.0 (7.94) | 8.9 (8.11) | 9.3 (9.20)
  Week 28: number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 | 7.7 (9.67) | 9.5 (8.22) | 7.2 (7.73) | 12.3 (11.48) | 9.8 (10.02) | 11.7 (10.41)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | 7.4 (9.51) | 8.4 (8.25) | 7.3 (5.54) | 10.6 (11.36) | 9.6 (6.48) | 11.3 (11.23)
  Week 44: number analyzed (Participants) | 47 | 54 | 10 | 12 | 27 | 28
  Week 44 | 7.8 (9.00) | 10.0 (9.52) | 7.9 (5.07) | 13.1 (11.10) | 7.7 (7.89) | 11.8 (11.35)
  Week 52: number analyzed (Participants) | 43 | 52 | 10 | 12 | 24 | 26
  Week 52 | 7.8 (8.54) | 10.4 (9.86) | 9.4 (9.01) | 12.3 (12.74) | 10.5 (8.91) | 10.5 (10.62)

22. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey (SF-36) Version 2, Acute at Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The SF-36 version 2 (Acute version) is a 36-item generic health status measure. It measures 8 general health concepts or domains: Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE), and Mental Health (MH). These 8 domains can also be summarized as physical and mental component scores. The summary component scores, Physical Component Summary (PCS) and Mental Component Summary (MCS), are based on a normalized sum of the 8 scale scores PF, RP, BP, GH, VT, SF, RE, and MH. All domains and summary components are scored such that a higher score indicates a higher functioning or health level. The minimum and maximum scores of the PCS Score are 22 and 59 respectively. The minimum and maximum scores of the MCS Score are 11 and 62 respectively.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Units on a scale
  Week 4 (Physical Component Summary Score): number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 4 (Physical Component Summary Score) | 3.29 (7.092) | 4.24 (7.602) | 2.59 (5.263) | 1.01 (3.944) | 1.66 (5.845) | 2.64 (6.299)
  Week 8 (Physical Component Summary Score): number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 (Physical Component Summary Score) | 4.21 (8.297) | 5.97 (8.261) | 5.53 (9.387) | 2.47 (3.675) | 2.57 (6.457) | 3.04 (5.529)
  Week 12 (Physical Component Summary Score): number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 (Physical Component Summary Score) | 4.09 (8.403) | 4.86 (9.010) | 7.28 (7.232) | 2.29 (4.283) | 2.22 (6.205) | 3.07 (7.330)
  Week 16 (Physical Component Summary Score): number analyzed (Participants) | 57 | 57 | 14 | 13 | 31 | 31
  Week 16 (Physical Component Summary Score) | 5.40 (8.239) | 7.27 (8.627) | 6.97 (7.223) | 5.07 (4.763) | 2.36 (6.842) | 1.79 (6.101)
  Week 20 (Physical Component Summary Score): number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 (Physical Component Summary Score) | 4.75 (8.579) | 8.84 (8.231) | 9.53 (8.434) | 2.03 (6.756) | 6.14 (7.513) | 6.25 (8.447)
  Week 28 (Physical Component Summary Score): number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 (Physical Component Summary Score) | 6.16 (8.691) | 9.06 (9.597) | 9.42 (7.751) | 7.84 (7.127) | 5.67 (7.933) | 9.22 (8.890)
  Week 36 (Physical Component Summary Score): number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 (Physical Component Summary Score) | 6.58 (9.510) | 7.75 (9.223) | 9.08 (9.789) | 6.44 (7.245) | 5.96 (6.738) | 9.41 (8.940)
  Week 44 (Physical Component Summary Score): number analyzed (Participants) | 47 | 54 | 10 | 12 | 27 | 28
  Week 44 (Physical Component Summary Score) | 6.67 (9.541) | 9.23 (9.477) | 8.44 (9.527) | 7.13 (6.759) | 6.00 (6.937) | 9.18 (8.199)
  Week 52 (Physical Component Summary Score): number analyzed (Participants) | 43 | 52 | 10 | 12 | 24 | 26
  Week 52 (Physical Component Summary Score) | 6.52 (9.818) | 9.98 (9.150) | 9.55 (9.536) | 6.64 (7.925) | 7.21 (8.130) | 9.84 (9.347)
  Week 4 (Mental Component Summary Score): number analyzed (Participants) | 59 | 58 | 16 | 15 | 33 | 33
  Week 4 (Mental Component Summary Score) | -0.28 (10.643) | 3.79 (9.139) | 1.24 (5.426) | 3.99 (10.723) | 0.45 (7.539) | -1.09 (9.805)
  Week 8 (Mental Component Summary Score): number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 (Mental Component Summary Score) | 0.84 (9.810) | 2.84 (10.894) | -2.05 (10.553) | 6.91 (10.450) | 0.29 (10.253) | 0.75 (8.880)
  Week 12 (Mental Component Summary Score): number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 (Mental Component Summary Score) | 0.85 (9.860) | 4.99 (10.307) | 0.78 (8.488) | 5.15 (13.189) | 1.37 (11.261) | 1.50 (9.640)
  Week 16 (Mental Component Summary Score): number analyzed (Participants) | 57 | 57 | 14 | 13 | 31 | 31
  Week 16 (Mental Component Summary Score) | 2.25 (10.848) | 2.12 (11.369) | 1.01 (6.995) | 4.78 (10.930) | 2.83 (8.459) | 3.03 (9.824)
  Week 20 (Mental Component Summary Score): number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 (Mental Component Summary Score) | 2.44 (10.131) | 3.59 (10.763) | 2.76 (8.595) | 6.58 (10.796) | 4.99 (8.782) | 6.72 (8.781)
  Week 28 (Mental Component Summary Score): number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 (Mental Component Summary Score) | 3.85 (11.295) | 3.64 (11.004) | 3.54 (7.290) | 8.95 (12.914) | 6.08 (7.764) | 6.57 (9.590)
  Week 36 (Mental Component Summary Score): number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 (Mental Component Summary Score) | 3.98 (9.044) | 5.41 (11.649) | 4.74 (9.301) | 8.53 (14.210) | 6.58 (7.419) | 5.47 (10.182)
  Week 44 (Mental Component Summary Score): number analyzed (Participants) | 47 | 54 | 10 | 12 | 27 | 28
  Week 44 (Mental Component Summary Score) | 5.14 (9.745) | 4.43 (13.601) | 4.29 (10.641) | 7.70 (13.606) | 6.33 (7.785) | 4.98 (10.544)
  Week 52 (Mental Component Summary Score): number analyzed (Participants) | 43 | 52 | 10 | 12 | 24 | 26
  Week 52 (Mental Component Summary Score) | 4.12 (10.023) | 4.33 (13.303) | 3.63 (10.656) | 8.69 (16.192) | 5.68 (8.783) | 4.35 (10.770)

23. Secondary Outcome: Percentage of Participants Achieving Minimal Disease Activity (MDA) at Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: A psoriatic arthritis participant was defined as having MDA response when 5 of the 7 following criteria were met: 1) tender joint count ≤1; 2) swollen joint count ≤1; 3) Psoriasis Area and Severity Index (quantifying the severity of a participant's psoriasis based on both lesion severity and the percentage of body surface area affected) score ≤1 or Body Surface Area (assessment of body surface area involved in psoriasis) ≤3%; 4) Patient's Assessment of Arthritis Pain (assessment of the patient's level of pain using a horizontal 100 mm visual analog scale) ≤15 mm; 5) Patient's Global Arthritis Assessment (patient's overall assessment of how the arthritis was doing by a 100 mm visual analog scale) ≤20 mm; 6) Health Assessment Questionnaire - Disability Index (assessment of the degree of difficulty a patient experienced) score ≤0.5; 7) tender entheseal points (assessment of tenderness using Leed's Enthesitis Index) ≤1.
Time Frame: Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Percentage of participants
  Week 4 | 8.33 [1.34 to 15.33] | 8.33 [1.34 to 15.33] | 6.25 [0.00 to 18.11] | 3.13 [0.00 to 11.65] | 1.43 [0.00 to 5.36] | 3.03 [0.00 to 8.88]
  Week 8 | 26.67 [15.48 to 37.86] | 21.67 [11.24 to 32.09] | 18.75 [0.00 to 37.87] | 6.67 [0.00 to 19.29] | 5.88 [0.00 to 13.79] | 12.12 [0.99 to 23.26]
  Week 12 | 31.67 [19.90 to 43.44] | 25.00 [14.04 to 35.96] | 18.75 [0.00 to 37.87] | 20.00 [0.00 to 40.24] | 5.88 [0.00 to 13.79] | 12.12 [0.99 to 23.26]
  Week 16: number analyzed (Participants) | 59 | 60 | 16 | 15 | 34 | 33
  Week 16 | 35.59 [23.38 to 47.81] | 35.00 [22.93 to 47.07] | 18.75 [0.00 to 37.87] | 20.00 [0.00 to 40.24] | 2.94 [0.00 to 8.62] | 3.03 [0.00 to 8.88]
  Week 20 | 45.00 [32.41 to 57.59] | 38.33 [26.03 to 50.64] | 25.00 [3.78 to 46.22] | 26.67 [4.29 to 49.05] | 29.41 [14.10 to 44.73] | 24.24 [9.62 to 38.86]
  Week 28 | 43.33 [30.79 to 55.87] | 46.67 [34.04 to 59.29] | 31.25 [8.54 to 53.96] | 33.33 [9.48 to 57.19] | 32.35 [16.63 to 48.08] | 45.45 [28.47 to 62.44]
  Week 36 | 43.33 [30.79 to 55.87] | 43.33 [30.79 to 55.87] | 50.00 [25.50 to 74.50] | 60.00 [35.21 to 84.79] | 29.41 [14.10 to 44.73] | 57.58 [40.71 to 74.44]
  Week 44 | 53.33 [40.71 to 65.96] | 50.00 [37.35 to 62.65] | 31.25 [8.54 to 53.96] | 46.67 [21.42 to 71.91] | 32.35 [16.63 to 48.08] | 51.52 [34.46 to 68.57]
  Week 52 | 46.67 [34.04 to 59.29] | 48.33 [35.69 to 60.98] | 31.25 [8.54 to 53.96] | 40.00 [15.21 to 64.79] | 41.18 [24.63 to 57.72] | 45.45 [28.47 to 62.44]

24. Secondary Outcome: Percentage of Participants Achieving Very Low Disease Activity (VLDA) Response at Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: A participant was in VLDA when all the 7 following criteria were met: 1) tender joint count ≤1; 2) swollen joint count ≤1; 3) Psoriasis Area and Severity Index (quantifying the severity of a participant's psoriasis based on both lesion severity and the percentage of body surface area affected) score ≤1 or Body Surface Area (assessment of body surface area involved in psoriasis) ≤3%; 4) Patient's Assessment of Arthritis Pain (assessment of the patient's level of pain using a horizontal 100 mm visual analog scale) ≤15 mm; 5) Patient's Global Arthritis Assessment (patient's overall assessment of how the arthritis was doing by a 100 mm visual analog scale) ≤20 mm; 6) Health Assessment Questionnaire - Disability Index (assessment of the degree of difficulty a patient experienced) score ≤0.5; 7) tender entheseal points (assessment of tenderness using Leed's Enthesitis Index) ≤1.
Time Frame: Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Percentage of participants
  Week 4 | 0.82 [0.00 to 3.08] | 0.82 [0.00 to 3.08] | 2.94 [0.00 to 10.97] | 3.13 [0.00 to 11.65] | 1.43 [0.00 to 5.36] | 1.47 [0.00 to 5.52]
  Week 8 | 1.67 [0.00 to 4.91] | 1.67 [0.00 to 4.91] | 2.94 [0.00 to 10.97] | 3.13 [0.00 to 11.65] | 1.43 [0.00 to 5.36] | 1.47 [0.00 to 5.52]
  Week 12 | 0.82 [0.00 to 3.08] | 3.33 [0.00 to 7.88] | 2.94 [0.00 to 10.97] | 3.13 [0.00 to 11.65] | 1.43 [0.00 to 5.36] | 1.47 [0.00 to 5.52]
  Week 16: number analyzed (Participants) | 59 | 60 | 16 | 15 | 34 | 33
  Week 16 | 3.39 [0.00 to 8.01] | 5.00 [0.00 to 10.51] | 6.25 [0.00 to 18.11] | 3.13 [0.00 to 11.65] | 1.43 [0.00 to 5.36] | 1.47 [0.00 to 5.52]
  Week 20 | 6.67 [0.35 to 12.98] | 11.67 [3.54 to 19.79] | 12.50 [0.00 to 28.70] | 13.33 [0.00 to 30.54] | 2.94 [0.00 to 8.62] | 1.47 [0.00 to 5.52]
  Week 28 | 10.00 [2.41 to 17.59] | 10.00 [2.41 to 17.59] | 12.50 [0.00 to 28.70] | 6.67 [0.00 to 19.29] | 8.82 [0.00 to 18.36] | 6.06 [0.00 to 14.20]
  Week 36 | 15.00 [5.97 to 24.03] | 15.00 [5.97 to 24.03] | 12.50 [0.00 to 28.70] | 6.67 [0.00 to 19.29] | 5.88 [0.00 to 13.79] | 12.12 [0.99 to 23.26]
  Week 44 | 15.00 [5.97 to 24.03] | 16.67 [7.24 to 26.10] | 18.75 [0.00 to 37.87] | 20.00 [0.00 to 40.24] | 14.71 [2.80 to 26.61] | 15.15 [2.92 to 27.38]
  Week 52 | 20.00 [9.88 to 30.12] | 16.67 [7.24 to 26.10] | 25.00 [3.78 to 46.22] | 20.00 [0.00 to 40.24] | 11.76 [0.93 to 22.59] | 18.18 [5.02 to 31.34]

25. Secondary Outcome: Change From Baseline in the Disease Activity Index for Reactive Arthritis/PsA (DAREA/DAPSA) at Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: DAREA/DAPSA is a composite instrument to assess peripheral joint involvement that is based upon numerical summation of 5 variables of disease activity: tender/painful joint count + swollen joint count (using SJC66/ TJC68 assessments), Patient's Global Assessment of Arthritis (PtGA in cm), Patient's Assessment of Arthritis Pain (PAIN in cm) and C-reactive protein (CRP) (in mg/dL). Since DAREA reflects domains found important in PsA, it has been proposed to serve as a Disease Activity Index for Psoriatic Arthritis (DAPSA). DAREA/DAPSA was calculated as follows: DAREA/DAPSA= SJC66 + TJC68 + PtGA + PAIN + CRP. A negative change from baseline represents improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: "Overall Number of Participants Analyzed" included all the participants in the evaluable population (participants who were randomized to the study and received at least one dose of the randomized study treatment) with baseline DAREA/DAPSA. "Number Analyzed" included participants available in the evaluable population at each specified treatment timepoints with baseline DAREA/DAPSA.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Units on a scale
  Week 4: number analyzed (Participants) | 58 | 57 | 16 | 15 | 33 | 33
  Week 4 | -14.05 (11.826) | -13.99 (10.166) | -14.15 (14.294) | -9.81 (13.841) | -7.11 (8.738) | -9.08 (12.074)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | -20.36 (11.211) | -17.55 (11.664) | -19.19 (11.720) | -14.33 (15.143) | -12.46 (12.905) | -10.98 (15.222)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | -21.93 (12.582) | -20.91 (11.985) | -24.91 (15.556) | -17.77 (18.471) | -14.68 (12.943) | -13.04 (15.072)
  Week 16: number analyzed (Participants) | 56 | 57 | 14 | 13 | 30 | 31
  Week 16 | -25.15 (12.582) | -23.55 (12.040) | -26.65 (16.982) | -25.89 (18.513) | -15.83 (12.918) | -14.45 (15.150)
  Week 20: number analyzed (Participants) | 54 | 56 | 13 | 13 | 31 | 31
  Week 20 | -26.75 (13.625) | -25.24 (12.152) | -30.63 (17.150) | -27.01 (22.334) | -23.53 (13.606) | -23.63 (13.640)
  Week 28: number analyzed (Participants) | 52 | 56 | 13 | 13 | 29 | 30
  Week 28 | -27.13 (12.807) | -25.38 (13.129) | -32.63 (18.437) | -31.41 (22.145) | -23.54 (12.375) | -27.55 (14.831)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | -27.21 (14.456) | -25.84 (13.170) | -34.98 (19.857) | -31.53 (24.046) | -25.57 (11.445) | -28.22 (15.793)
  Week 44: number analyzed (Participants) | 46 | 54 | 10 | 12 | 27 | 28
  Week 44 | -28.39 (14.445) | -27.54 (12.744) | -36.61 (14.597) | -30.22 (27.532) | -26.43 (10.880) | -29.59 (15.962)
  Week 52: number analyzed (Participants) | 41 | 50 | 10 | 12 | 23 | 26
  Week 52 | -28.56 (15.578) | -27.40 (13.429) | -37.81 (14.251) | -30.32 (22.795) | -26.45 (11.114) | -28.95 (17.706)

26. Secondary Outcome: Percentage of Participants Achieving the Psoriatic Arthritis Response Criteria (PsARC) at Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: The PsARC response was defined as improvement in two of the following 4 criteria, one of which must be joint pain or swelling, without worsening in any measure: (1) ≥20% improvement in Physician's Global Assessment of Arthritis (a horizontal visual analog scale measure of the physician's assessment of the patient's current disease activity); (2) ≥20% improvement in Patient's Global Assessment of Arthritis (the patient's overall assessment of how the arthritis was doing by a visual analog scale); (3) ≥30% improvement in tender joint count (68); and (4) ≥30% improvement in swollen joint count.
Time Frame: Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: "Overall Number of Participants Analyzed" indicated the evaluable population and included all participants who were randomized to the study and received at least one dose of the randomized study treatment. "Number Analyzed" included participants available in the evaluable population at each specified treatment timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Percentage of participants
  Week 4 | 50.00 [37.35 to 62.65] | 55.00 [42.41 to 67.59] | 50.00 [25.50 to 74.50] | 40.00 [15.21 to 64.79] | 26.47 [11.64 to 41.30] | 21.21 [7.26 to 35.16]
  Week 8 | 66.67 [54.74 to 78.59] | 60.00 [47.60 to 72.40] | 56.25 [31.94 to 80.56] | 40.00 [15.21 to 64.79] | 38.24 [21.90 to 54.57] | 45.45 [28.47 to 62.44]
  Week 12 | 66.67 [54.74 to 78.59] | 75.00 [64.04 to 85.96] | 62.50 [38.78 to 86.22] | 60.00 [35.21 to 84.79] | 52.94 [36.16 to 69.72] | 45.45 [28.47 to 62.44]
  Week 16: number analyzed (Participants) | 59 | 60 | 16 | 15 | 34 | 33
  Week 16 | 83.05 [73.48 to 92.62] | 75.00 [64.04 to 85.96] | 62.50 [38.78 to 86.22] | 66.67 [42.81 to 90.52] | 50.00 [33.19 to 66.81] | 48.48 [31.43 to 65.54]
  Week 20 | 78.33 [67.91 to 88.76] | 81.67 [71.88 to 91.46] | 56.25 [31.94 to 80.56] | 60.00 [35.21 to 84.79] | 70.59 [55.27 to 85.90] | 72.73 [57.53 to 87.92]
  Week 28 | 81.67 [71.88 to 91.46] | 80.00 [69.88 to 90.12] | 68.75 [46.04 to 91.46] | 73.33 [50.95 to 95.71] | 73.53 [58.70 to 88.36] | 75.76 [61.14 to 90.38]
  Week 36 | 66.67 [54.74 to 78.59] | 75.00 [64.04 to 85.96] | 68.75 [46.04 to 91.46] | 80.00 [59.76 to 100.00] | 67.65 [51.92 to 83.37] | 84.85 [72.62 to 97.08]
  Week 44 | 66.67 [54.74 to 78.59] | 78.33 [67.91 to 88.76] | 56.25 [31.94 to 80.56] | 73.33 [50.95 to 95.71] | 58.82 [42.28 to 75.37] | 75.76 [61.14 to 90.38]
  Week 52 | 58.33 [45.86 to 70.81] | 70.00 [58.40 to 81.60] | 56.25 [31.94 to 80.56] | 66.67 [42.81 to 90.52] | 64.71 [48.64 to 80.77] | 66.67 [50.58 to 82.75]

27. Secondary Outcome: Change From Baseline in the Psoriatic Arthritis Disease Activity Score (PASDAS) at Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Description: PASDAS is a composite psoriatic arthritis disease activity score that includes the following components: patient's global joint and skin assessment (visual analog scale in mm), physician's global psoriatic arthritis assessment (visual analog scale in mm), swollen (66 joints) and tender joint counts (68 joints), Leeds Enthesitis Index score, tender dactylitic digit score, physical component summary score (PCS) of Short Form 36 Health Survey and C-reactive protein (mg/L). Any missing component would result in PASDAS as missing. A higher PASDAS score indicates a higher disease activity.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 28, 36, 44 and 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Units on a scale
  Week 4: number analyzed (Participants) | 59 | 57 | 16 | 15 | 33 | 33
  Week 4 | -1.22 (1.119) | -1.31 (1.090) | -0.94 (0.957) | -0.65 (0.653) | -0.56 (0.655) | -0.54 (0.897)
  Week 8: number analyzed (Participants) | 58 | 57 | 16 | 14 | 32 | 33
  Week 8 | -1.79 (1.295) | -1.65 (1.262) | -1.37 (1.127) | -1.14 (1.122) | -1.02 (0.988) | -0.67 (1.045)
  Week 12: number analyzed (Participants) | 58 | 57 | 14 | 14 | 31 | 33
  Week 12 | -2.10 (1.380) | -1.93 (1.278) | -1.67 (0.996) | -1.61 (1.106) | -1.04 (1.101) | -0.80 (1.158)
  Week 16: number analyzed (Participants) | 56 | 57 | 14 | 13 | 30 | 31
  Week 16 | -2.31 (1.302) | -2.20 (1.354) | -1.87 (1.024) | -2.18 (1.286) | -1.08 (1.127) | -0.90 (1.193)
  Week 20: number analyzed (Participants) | 55 | 56 | 13 | 13 | 31 | 31
  Week 20 | -2.48 (1.338) | -2.48 (1.474) | -2.49 (1.199) | -2.18 (1.441) | -2.37 (1.202) | -2.10 (1.367)
  Week 28: number analyzed (Participants) | 52 | 55 | 13 | 13 | 29 | 30
  Week 28 | -2.62 (1.354) | -2.60 (1.642) | -2.90 (1.279) | -3.18 (1.484) | -2.48 (1.181) | -2.81 (1.302)
  Week 36: number analyzed (Participants) | 49 | 56 | 13 | 13 | 27 | 29
  Week 36 | -2.73 (1.509) | -2.59 (1.644) | -3.08 (1.539) | -2.97 (1.550) | -2.69 (1.043) | -2.96 (1.425)
  Week 44: number analyzed (Participants) | 46 | 54 | 10 | 12 | 27 | 28
  Week 44 | -2.95 (1.421) | -2.85 (1.637) | -3.25 (0.819) | -3.23 (1.833) | -2.73 (1.157) | -3.23 (1.508)
  Week 52: number analyzed (Participants) | 41 | 50 | 10 | 12 | 23 | 26
  Week 52 | -3.03 (1.487) | -2.98 (1.568) | -3.36 (0.826) | -3.14 (1.461) | -2.84 (1.399) | -3.07 (1.775)

28. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) From Baseline (Day 1) Through Week 56 (All Causalities)
Description: Treatment-emergent AEs are those with initial onset or that worsen in severity after the first dose of the study medication. All AEs in the table below were treatment-emergent AEs. An SAE is any untoward medical occurrence at any dose that: results in death; is life threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect; or that is considered to be an important medical event that may jeopardize the participant or may require intervention to prevent one of the other AE outcomes. Severe AEs were defined as AEs that interfered significantly with participant's usual function. Both SAEs and severe AEs were according to the investigator's assessment.
Time Frame: Baseline (Day 1) through Week 56
Population: All participants who received at least one dose of the randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Participants
  Participants with AEs | 46 | 45 | 10 | 10 | 24 | 25
  Participants with SAEs | 1 | 8 | 0 | 0 | 1 | 2
  Participants with severe AEs | 1 | 6 | 0 | 0 | 1 | 2
  Participants with dose reduction or temporary discontinuation due to AEs | 18 | 14 | 4 | 3 | 4 | 8

29. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) From Baseline (Day 1) Through Week 56 (Treatment-related)
Description: Treatment-emergent AEs are those with initial onset or that worsen in severity after the first dose of the study medication. All AEs in the table below were treatment-emergent AEs. An SAE is any untoward medical occurrence at any dose that: results in death; is life threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect; or that is considered to be an important medical event that may jeopardize the participant or may require intervention to prevent one of the other AE outcomes. Severe AEs were defined as AEs that interfered significantly with participant's usual function. Both SAEs and severe AEs were according to the investigator's assessment. Treatment-related AEs were also determined by the investigator.
Time Frame: Baseline (Day 1) through Week 56
Population: All participants who received at least one dose of the randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Participants
  Participants with AEs | 17 | 15 | 6 | 2 | 11 | 10
  Participants with SAEs | 0 | 1 | 0 | 0 | 1 | 1
  Participants with severe AEs | 0 | 1 | 0 | 0 | 1 | 1
  Participants with dose reduction or temporary discontinuation due to AEs | 8 | 5 | 4 | 1 | 1 | 3

30. Secondary Outcome: Number of Participants Who Discontinued From Study Due to Treatment-emergent AEs From Baseline (Day 1) Through Week 56
Description: An AE is any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Treatment-emergent AEs were those with initial onset or that worsen in severity after the first dose of the study medication.
Time Frame: Baseline (Day 1) through Week 56
Population: All participants who received at least one dose of the randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
Number analyzed (Participants) | 60 | 60 | 16 | 15 | 34 | 33
Participants
  Otitis media acute | 0 | 1 | 0 | 0 | 0 | 0
  Upper respiratory tract infection | 0 | 0 | 0 | 0 | 0 | 1
  Psoriasis | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From the time the participants received the study treatment up to 28 days after the last treatment administration (approximately 56 weeks).
Description: The analysis of adverse events included all participants who received at least 1 dose of the randomized study treatment. The participants were analyzed according to the study treatment they actually received.
Arm/Group | PF-06700841 60 mg QD -> PF-06700841 60 mg QD | PF-06700841 30 mg QD -> PF-06700841 30 mg QD | PF-06700841 10 mg QD -> PF-06700841 60 mg QD | PF-06700841 10 mg QD -> PF-06700841 30 mg QD | Placebo -> PF-06700841 60 mg QD | Placebo -> PF-06700841 30 mg QD
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/16 | 0/15 | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/60 | 8/60 | 0/16 | 0/15 | 1/34 | 2/33
Other Adverse Events (participants affected / at risk) | 37/60 | 34/60 | 10/16 | 10/15 | 18/34 | 20/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06700841 60 mg QD -> PF-06700841 60 mg QD (N=60) | PF-06700841 30 mg QD -> PF-06700841 30 mg QD (N=60) | PF-06700841 10 mg QD -> PF-06700841 60 mg QD (N=16) | PF-06700841 10 mg QD -> PF-06700841 30 mg QD (N=15) | Placebo -> PF-06700841 60 mg QD (N=34) | Placebo -> PF-06700841 30 mg QD (N=33)
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06700841 60 mg QD -> PF-06700841 60 mg QD (N=60) | PF-06700841 30 mg QD -> PF-06700841 30 mg QD (N=60) | PF-06700841 10 mg QD -> PF-06700841 60 mg QD (N=16) | PF-06700841 10 mg QD -> PF-06700841 30 mg QD (N=15) | Placebo -> PF-06700841 60 mg QD (N=34) | Placebo -> PF-06700841 30 mg QD (N=33)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 3 | 1
Fatigue (General disorders) | 3 | 1 | 1 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 0 | 1 | 2 | 1 | 1
COVID-19 (Infections and infestations) | 1 | 2 | 0 | 1 | 1 | 2
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 8 | 5 | 0 | 2 | 1 | 4
Oral herpes (Infections and infestations) | 2 | 2 | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 5 | 0 | 0 | 2 | 3
Urinary tract infection (Infections and infestations) | 4 | 4 | 1 | 1 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 7 | 1 | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 0 | 1 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 4 | 4 | 1 | 0 | 1 | 2
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 1 | 0 | 2 | 0
Hepatic enzyme increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 1 | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 1
Headache (Nervous system disorders) | 5 | 4 | 2 | 1 | 1 | 3
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 5 | 2 | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT03963401/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT03963401/SAP_001.pdf